CLINICAL TRIAL: NCT02783300
Title: A Phase I, Open-label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of GSK3326595 in Subjects With Solid Tumors and Non-Hodgkin's Lymphoma
Brief Title: An Open-label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of GSK3326595 in Participants With Solid Tumors and Non-Hodgkin's Lymphoma
Acronym: Meteor 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 204653; 2016-000278-39 (EudraCT Number)
Record Dates: First submitted 2016-04-11; First posted 2016-05-26 (Estimated); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Neoplasms
Keywords: GSK3326595; Solid tumor; Non-Hodgkin's lymphoma (NHL); Urinary tract cancer; Dose escalation; Adenoid cystic carcinoma (ACC); Non small-cell lung cancer (NSCLC); Squamous cell carcinoma of the head and neck (HNSCC); Melanoma
MeSH Terms: conditions — Neoplasms; Lymphoma, Non-Hodgkin; Urologic Neoplasms; Carcinoma, Adenoid Cystic; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Melanoma | interventions — GSK-3326595; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This will be a three-part study where Part 1 is dose escalation, including assessment of Food Effect and Relative Bioavailability, Part 2 is disease specific expansion cohorts to better characterize the clinical activity and safety profile of GSK3326595 and Part 3 is dose determination of GSK3326595 in combination with pembrolizumab.
Masking Description: This is an open label study.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: Dose Escalation, Food effect and Relative Bioavailability of Capsule formulation to Tablet (Experimental): Participants will receive escalating doses of GSK3326595 until the maximum tolerated dose level is reached. The recommended phase 2 dose (RP2D) will be determined. Participants will be dosed in a fed (high-fat, high-calorie meal) and fasted state to determine the effect of food on bioavailability of GSK3326595, and will be dosed with tablet and capsule to compare two formulations of GSK3326595 (capsule versus tablet).
  Interventions: Drug: GSK3326595
- Part 2: Disease-Specific Expansion cohort (Experimental): Participants with triple-negative breast cancer (TNBC), metastatic transitional cell carcinoma of the urinary system (mTCC), Grade IV anaplastic astrocytoma (glioblastoma multiforme [GBM]), non-Hodgkin's lymphoma (NHL), adenoid cystic carcinoma (ACC), hormone receptor-positive adenocarcinoma of the breast (ER+BC), human papillomavirus (HPV)-positive solid tumors of any histology, and p53-wild type non-small cell lung cancer (NSCLC) will be administered GSK3326595 at the recommended phase 2 dose (RP2D) as determined in Part 1.
  Interventions: Drug: GSK3326595
- Part 3: GSK3326595 in combination with pembrolizumab (Experimental): Participants with selected solid tumors will be administered GSK3326595 in combination with pembrolizumab as part of this dose determination study.
  Interventions: Drug: GSK3326595; Drug: Pembrolizumab

INTERVENTIONS:
Drug: GSK3326595 — GSK3326595 will be administered with and without food, in tablet and capsule formulation.
Drug: Pembrolizumab — Pembrolizumab will be administered.
  Arms: Part 3: GSK3326595 in combination with pembrolizumab

SUMMARY:
This first time in human (FTIH) open-label, dose escalation study will assess the safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of GSK3326595 in participants with advanced or recurrent solid tumors, as well as clinical activity in participants with a subset of solid tumors and non-Hodgkin's lymphoma (NHL).

ELIGIBILITY:
Inclusion criteria:

* Males and females greater than or equal to (>=)18 years of age (at the time consent is obtained)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 or 2
* Diagnosis of non-resectable or metastatic solid malignancy (as defined in the protocol) or NHL
* Presence of evaluable disease
* Adequate organ function (as defined in the protocol)
* Reproductive criteria (as defined in the protocol).

Exclusion Criteria:

* Malignancy attributed to prior solid organ transplant
* Leptomeningeal disease, spinal cord compression, or brain metastases that require immediate central nervous system (CNS)-specific treatment in the opinion of the Investigator (for example [e.g.], for symptomatic disease)
* History of a second malignancy, excluding non-melanoma skin cell cancer within the last three years
* Evidence of severe or uncontrolled systemic diseases, or serious and/or pre-existing medical or other condition that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator
* Any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.
* Select cardiac abnormalities (as defined in the protocol)
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* History of optic nerve neuropathy or neuritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (6):
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
- France (3):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Villejuif
- Netherlands (3):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD): Participant with relapsed and/or refractory solid tumors received 12.5 mg GSK3326595 capsules orally once a day until the maximally tolerated dose (MTD) was reached.
- Part 1: GSK3326595 25mg QD: Participant with relapsed and/or refractory solid tumors received 25 mg GSK3326595 capsules orally once a day until the MTD was reached.
- Part 1: GSK3326595 50mg QD: Participant with relapsed and/or refractory solid tumors received 50 mg GSK3326595 capsules orally once a day until the MTD was reached.
- Part 1: GSK3326595 100mg QD: Participant with relapsed and/or refractory solid tumors received 100 mg GSK3326595 capsules orally once a day until the MTD was reached.
- Part 1: GSK3326595 200mg QD: Participant with relapsed and/or refractory solid tumors received 200 mg GSK3326595 capsules orally once a day until the MTD was reached.
- Part 1: GSK3326595 300mg QD: Participant with relapsed and/or refractory solid tumors received 300 mg GSK3326595 capsules orally once a day until the MTD was reached.
- Part 1: GSK3326595 400mg QD: Participant with relapsed and/or refractory solid tumors received 400 mg GSK3326595 capsules orally once a day.
- Part 1: GSK3326595 600mg QD: Participant with relapsed and/or refractory solid tumors received 600 mg GSK3326595 capsules orally once a day.
- Part 1: GSK3326595 50mg Twice Daily (BID): Participant with relapsed and/or refractory solid tumors received 50 mg GSK3326595 capsules twice a day.
- Part 1: GSK3326595 100mg BID: Participant with relapsed and/or refractory solid tumors received 100 mg GSK3326595 capsules twice a day.
- Part 1: GSK3326595 150mg BID: Participant with relapsed and/or refractory solid tumors received 150 mg GSK3326595 capsules twice a day.
- Part 1: GSK3326595 200mg BID: Participant with relapsed and/or refractory solid tumors received 200 mg GSK3326595 capsules twice a day.
- Part 1: GSK3326595 300mg QD (Food Effect): Participant with relapsed and/or refractory solid tumors received 300 mg GSK3326595 once a day (QD) tablet/capsule under fasting conditions, with no food or antacids for 1 h before and 2 h after each dose OR under fed condition with recommended high fat, high calorie breakfast 30 minutes prior to administration of GSK3326595.
- Part 2: GSK3326595 400mg (TNBC): Participant with triple-negative breast cancer (TNBC) received 400 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 400mg (mTCC): Participant with metastatic transitional cell carcinoma of the urinary system (mTCC) received 400 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 400mg (GBM): Participant with Grade IV anaplastic astrocytoma (glioblastoma multiforme [GBM]) received 400 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 400mg (ER+BC): Participant with hormone receptor-positive adenocarcinoma of the breast (ER+BC) received 400 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 400mg (HPV+): Participant with human papillomavirus (HPV)-positive solid tumors received 400 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 400mg (ACC): Participant with adenoid cystic carcinoma (ACC) received 400 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 300mg (ACC): Participant with ACC received 300 mg GSK3326595 tablets orally once a day.
- Part 2: GSK3326595 400mg (NHL P53 Mutant): Participant with non-Hodgkin's lymphoma (NHL) P53 Mutant received 400 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 300mg (NHL P53 Mutant): Participant with NHL P53 Mutant received 300 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 400mg (NHL P53 Wild Type): Participant with NHL P53 Wild Type received 400 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 300mg (NHL P53 Wild Type): Participant with NHL P53 Wild Type received 300 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 400mg (NHL P53 Unknown): Participant with NHL P53 Unknown received 400 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 300mg (NSCLC): Participant with non-small cell lung cancer (NSCLC) received 300 mg GSK3326595 capsules orally once a day.
- Part 3: GSK3326595 100mg + Pembrolizumab 200mg: Participant with NSCLC, mTCC, melanoma, and HNSCC received 100 mg GSK3326595 capsules in combination with 200 mg Pembrolizumab orally once a day.
Period: Part 1- Dose Escalation Phase
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect) | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC) | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Started | 1 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 0 | 7 | 3 | 13 | 3 | 1 | 6 | 6 | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 1 | 0 | 6 | 0 | 0 | 1 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Site Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator discretion | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2- Disease-specific Expansion Phase
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect) | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC) | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 16 | 29 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 10 | 22 | 31 | 25 | 20 | 3 | 4 | 1 | 5 | 1 | 7 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 7 | 6 | 3 | 14 | 13 | 2 | 1 | 3 | 1 | 4 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Site Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator site closed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 0 | 7 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator discretion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 3 | 3 | 1 | 3 | 5 | 1 | 1 | 2 | 1 | 3 | 4 | 0
Period: Part 3- Dose Determination Phase
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect) | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC) | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Investigator discretion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect) | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC) | Part 3: GSK3326595 100mg + Pembrolizumab 200mg | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15 | 22 | 16 | 29 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7 | 10 | 297
Age, Customized [Count of Participants; unit: Participants]
  18 - 84 Years | 1 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15 | 22 | 16 | 29 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7 | 10 | 297
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 5 | 2 | 8 | 2 | 1 | 2 | 1 | 2 | 7 | 22 | 5 | 6 | 37 | 23 | 16 | 11 | 2 | 1 | 3 | 1 | 2 | 2 | 4 | 167
  Male | 1 | 0 | 0 | 1 | 3 | 1 | 11 | 1 | 0 | 5 | 5 | 1 | 8 | 0 | 11 | 23 | 0 | 5 | 18 | 5 | 4 | 1 | 5 | 1 | 9 | 5 | 6 | 130
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race categories (with 0<n<11) are combined into 'Others' category to maintain participant confidentiality and privacy.
  Participants
    Others | 1 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15 | 22 | 16 | 28 | 37 | 28 | 34 | 15 | 6 | 2 | 8 | 2 | 11 | 7 | 9 | 294
    Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or is a congenital anomaly/birth defect, other situations which involved medical or scientific judgment or is associated with liver injury and impaired liver function. SAEs are subset of AEs. A summary of number of participants with any AEs and SAEs is presented. AEs were coded using the Medical Dictionary for Regulatory Affairs (MedDRA dictionary).
Time Frame: Up to 30 months
Population: All treated population included all participants who received at least one dose of GSK3326595.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
Participants
  Any AEs | 1 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
  Any SAEs | 0 | 0 | 0 | 0 | 4 | 1 | 10 | 1 | 0 | 2 | 3 | 3 | 6

2. Primary Outcome: Part 1: Number of Participants Withdrawn Due to AEs
Description: The data for number of participants withdrawn due to AEs have been presented.
Time Frame: Up to 30 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
Participants | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1

3. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT is considered to be clinically relevant AE by investigator if it met at least one of the criteria: Grade(G)3 neutropenia for >=5 days/G4 neutropenia of any duration, G3 or greater febrile neutropenia, G4 or greater anemia of any duration and thrombocytopenia, or G3 thrombocytopenia with bleeding, Alanine aminotransferase (ALT) >3x upper limit of normal (ULN)+bilirubin, >=2xULN or ALT between 3-5 X ULN with bilirubin < 2Xuln but with hepatitis symptoms/rash, G3 nausea/vomiting/diarrhea that does not improve within 72 hour, G4 or greater nausea/vomiting/diarrhea, G3 or greater hypertension, G3 or greater clinically significant non-hematologic toxicity per National Cancer Institute -- Common Terminology Criteria for Adverse Events (NCICTCAE), Inability to receive at least 80% of scheduled doses in the DLT observation period due to toxicity, G2 or higher toxicity that occurs beyond 21 days which in the judgment of the investigator and GSK Medical Monitor was considered to be a DLT.
Time Frame: Up to 21 days
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0

4. Primary Outcome: Part 1: Number of Participants With Dose Modifications of GSK3326595
Description: The number of participants who experienced any dose modifications (interruptions and reductions) of GSK3326595 have been presented.
Time Frame: Up to 30 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
Participants
  Dose interruptions | 1 | 1 | 1 | 1 | 5 | 3 | 18 | 2 | 0 | 5 | 4 | 2 | 14
  Dose reductions | 0 | 0 | 0 | 0 | 0 | 1 | 16 | 2 | 0 | 2 | 2 | 3 | 4

5. Primary Outcome: Part 1: Number of Participants With Worst Case Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for evaluation of clinical chemistry parameters. The summaries of worst-case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The number of participants with decreases to low, changes to normal or no changes from Baseline, and increases to high values have been presented. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Baseline (Day 1) and up to 30 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
Participants
  Alanine Aminotransferase, decreases to low | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 1 | 0 | 0 | 1 | 1 | 4
  Alanine Aminotransferase, changes to normal or no changes | 0 | 1 | 1 | 1 | 4 | 1 | 13 | 1 | 1 | 6 | 4 | 2 | 11
  Alanine Aminotransferase, increases to high | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 1 | 1 | 0 | 0
  Albumin, decreases to low | 1 | 1 | 1 | 1 | 4 | 1 | 12 | 1 | 0 | 2 | 5 | 1 | 7
  Albumin, changes to normal or no changes | 0 | 0 | 0 | 0 | 3 | 2 | 7 | 2 | 1 | 5 | 1 | 2 | 8
  Albumin, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase, changes to normal or no changes | 1 | 1 | 1 | 0 | 7 | 2 | 17 | 1 | 0 | 4 | 5 | 3 | 11
  Alkaline Phosphatase, increases to high | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 3 | 1 | 0 | 4
  Amylase, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2
  Amylase, changes to normal or no changes | 1 | 1 | 1 | 1 | 7 | 3 | 15 | 2 | 0 | 6 | 5 | 3 | 13
  Amylase, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0
  Aspartate Aminotransferase, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Aspartate Aminotransferase, changes to normal or no changes | 0 | 1 | 0 | 0 | 4 | 2 | 11 | 2 | 0 | 6 | 4 | 2 | 11
  Aspartate Aminotransferase, increases to high | 1 | 0 | 1 | 1 | 3 | 1 | 7 | 1 | 1 | 1 | 2 | 0 | 4
  Bilirubin, decreases to low | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Bilirubin, changes to normal or no changes | 1 | 1 | 1 | 1 | 5 | 2 | 13 | 2 | 0 | 3 | 4 | 2 | 13
  Bilirubin, increases to high | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 1 | 1 | 3 | 2 | 1 | 2
  Calcium, decreases to low | 1 | 0 | 0 | 0 | 3 | 2 | 12 | 1 | 1 | 4 | 3 | 1 | 7
  Calcium, changes to normal or no changes | 0 | 1 | 1 | 1 | 2 | 1 | 7 | 2 | 0 | 3 | 3 | 2 | 8
  Calcium, increases to high | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine, decreases to low | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2
  Creatinine, changes to normal or no changes | 1 | 1 | 0 | 0 | 6 | 3 | 16 | 3 | 1 | 6 | 4 | 3 | 11
  Creatinine, increases to high | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2
  Direct Bilirubin, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin, changes to normal or no changes | 1 | 1 | 1 | 1 | 3 | 2 | 11 | 2 | 0 | 2 | 4 | 1 | 9
  Direct Bilirubin, increases to high | 0 | 0 | 0 | 0 | 4 | 1 | 8 | 1 | 1 | 5 | 2 | 2 | 6
  Glucose, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Glucose, changes to normal or no changes | 1 | 1 | 1 | 1 | 6 | 3 | 9 | 1 | 0 | 4 | 5 | 0 | 11
  Glucose, increases to high | 0 | 0 | 0 | 0 | 1 | 0 | 10 | 1 | 1 | 3 | 1 | 3 | 3
  Lipase, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Lipase, changes to normal or no changes | 1 | 1 | 1 | 1 | 7 | 2 | 15 | 3 | 1 | 6 | 5 | 1 | 13
  Lipase, increases to high | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 2 | 0
  Potassium, decreases to low | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 5
  Potassium, changes to normal or no changes | 1 | 1 | 1 | 1 | 5 | 2 | 13 | 2 | 1 | 4 | 3 | 1 | 9
  Potassium, increases to high | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 2 | 3 | 2 | 1
  Protein, decreases to low | 1 | 0 | 0 | 0 | 3 | 0 | 12 | 1 | 0 | 4 | 4 | 1 | 6
  Protein, changes to normal or no changes | 0 | 1 | 1 | 1 | 4 | 3 | 6 | 2 | 1 | 3 | 2 | 2 | 8
  Protein, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Sodium, decreases to low | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 0 | 0 | 2 | 2 | 0 | 2
  Sodium, changes to normal or no changes | 1 | 1 | 1 | 1 | 3 | 2 | 14 | 3 | 1 | 5 | 3 | 3 | 11
  Sodium, increases to high | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Urea Nitrogen, decreases to low: number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 2 | 15 | 3 | 1 | 5 | 4 | 2 | 15
  Urea Nitrogen, decreases to low | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Urea Nitrogen, changes to normal or no changes: number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 2 | 15 | 3 | 1 | 5 | 4 | 2 | 15
  Urea Nitrogen, changes to normal or no changes | 1 | 1 | 1 | 0 | 3 | 2 | 9 | 2 | 0 | 2 | 2 | 2 | 11
  Urea Nitrogen, increases to high: number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 2 | 15 | 3 | 1 | 5 | 4 | 2 | 15
  Urea Nitrogen, increases to high | 0 | 0 | 0 | 0 | 4 | 0 | 6 | 1 | 0 | 3 | 2 | 0 | 3

6. Primary Outcome: Part 1: Number of Participants With Worst Case Change From Baseline in Hematology Parameters
Description: Blood samples were collected for evaluation of hematology parameters. The summaries of worst-case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with decreases to low, changes to normal or no changes from Baseline, and increases to high values have been presented. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Baseline (Day 1) and up to 30 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
Participants
  Basophils, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils, changes to normal or no changes | 1 | 1 | 1 | 1 | 6 | 2 | 19 | 3 | 1 | 7 | 6 | 2 | 15
  Basophils, increases to high | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Eosinophils, decreases to low | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Eosinophils, changes to normal or no changes | 1 | 0 | 1 | 1 | 5 | 3 | 16 | 3 | 1 | 6 | 6 | 0 | 14
  Eosinophils, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 0
  Mean Corpuscular Hemoglobin, decreases to low | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 6
  Mean Corpuscular Hemoglobin, changes to normal or no changes | 1 | 1 | 1 | 1 | 5 | 3 | 17 | 2 | 0 | 5 | 6 | 1 | 9
  Mean Corpuscular Hemoglobin, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
  Mean Corpuscular Volume, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Volume, changes to normal or no changes | 0 | 1 | 1 | 1 | 7 | 2 | 16 | 3 | 1 | 7 | 5 | 3 | 15
  Mean Corpuscular Volume, increases to high | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  Erythrocytes, decreases to low | 0 | 0 | 0 | 0 | 1 | 1 | 12 | 0 | 0 | 3 | 3 | 1 | 7
  Erythrocytes, changes to normal or no changes | 1 | 1 | 1 | 1 | 6 | 2 | 7 | 2 | 1 | 4 | 3 | 2 | 8
  Erythrocytes, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Hematocrit, decreases to low | 0 | 0 | 0 | 0 | 2 | 2 | 14 | 1 | 0 | 2 | 2 | 2 | 5
  Hematocrit, changes to normal or no changes | 1 | 1 | 1 | 1 | 5 | 1 | 5 | 2 | 1 | 5 | 4 | 1 | 10
  Hematocrit, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, decreases to low | 0 | 1 | 0 | 0 | 2 | 2 | 11 | 0 | 1 | 2 | 3 | 1 | 6
  Hemoglobin, changes to normal or no changes | 1 | 0 | 1 | 1 | 5 | 1 | 8 | 3 | 0 | 5 | 3 | 2 | 9
  Hemoglobin, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes, decreases to low | 1 | 0 | 0 | 0 | 2 | 2 | 8 | 1 | 0 | 4 | 1 | 2 | 8
  Leukocytes, changes to normal or no changes | 0 | 1 | 0 | 1 | 4 | 1 | 9 | 2 | 1 | 2 | 3 | 1 | 7
  Leukocytes, increases to high | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 2 | 1 | 0
  Lymphocytes, decreases to low | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 2 | 1 | 2 | 3 | 2 | 4
  Lymphocytes, changes to normal or no changes | 1 | 1 | 1 | 1 | 7 | 1 | 12 | 1 | 0 | 5 | 3 | 1 | 11
  Lymphocytes, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes, decreases to low | 0 | 1 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 0 | 1 | 0 | 0
  Monocytes, changes to normal or no changes | 1 | 0 | 1 | 1 | 4 | 1 | 10 | 3 | 1 | 7 | 3 | 2 | 12
  Monocytes, increases to high | 0 | 0 | 0 | 0 | 3 | 0 | 5 | 0 | 0 | 0 | 3 | 1 | 3
  Neutrophils, decreases to low | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 0 | 0 | 2 | 1 | 2 | 4
  Neutrophils, changes to normal or no changes | 1 | 1 | 0 | 1 | 4 | 1 | 9 | 1 | 1 | 3 | 2 | 1 | 10
  Neutrophils, increases to high | 0 | 0 | 1 | 0 | 3 | 0 | 5 | 2 | 0 | 2 | 3 | 1 | 2
  Neutrophils/ Leukocytes, decreases to low: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 1 | 8 | 3 | 1 | 3 | 2 | 1 | 8
  Neutrophils/ Leukocytes, decreases to low | 0 |  | 0 |  |  | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  Neutrophils/ Leukocytes, changes to normal or no changes: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 1 | 8 | 3 | 1 | 3 | 2 | 1 | 8
  Neutrophils/ Leukocytes, changes to normal or no changes | 1 |  | 1 |  |  | 1 | 5 | 2 | 1 | 2 | 0 | 1 | 6
  Neutrophils/ Leukocytes, increases to high: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 1 | 8 | 3 | 1 | 3 | 2 | 1 | 8
  Neutrophils/ Leukocytes, increases to high | 0 |  | 0 |  |  | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 2
  Platelets, decreases to low | 0 | 0 | 0 | 0 | 2 | 1 | 12 | 2 | 0 | 3 | 3 | 2 | 7
  Platelets, changes to normal or no changes | 1 | 1 | 1 | 1 | 4 | 2 | 4 | 1 | 1 | 4 | 3 | 0 | 7
  Platelets, increases to high | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 2
  Reticulocytes, decreases to low: number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
  Reticulocytes, decreases to low | 0 | 0 | 0 | 0 | 2 | 0 | 13 | 2 | 0 | 0 | 2 | 2 | 4
  Reticulocytes, changes to normal or no changes: number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
  Reticulocytes, changes to normal or no changes | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 0 | 1 | 3 | 2 | 1 | 4
  Reticulocytes, increases to high: number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
  Reticulocytes, increases to high | 0 | 0 | 0 | 0 | 2 | 2 | 13 | 2 | 0 | 4 | 2 | 1 | 8

7. Primary Outcome: Part 1: Number of Participants With Worst Case Change From Baseline in Coagulation Parameters
Description: Blood samples were collected for evaluation of coagulation parameters. The summaries of worst-case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v4.0. The number of participants with decreases to low, changes to normal or no changes from Baseline, and increases to high values have been presented. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Baseline (Day 1) and up to 30 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
Participants
  Partial Thromboplastin Time, decreases to low: number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 2 | 15 | 3 | 1 | 5 | 4 | 2 | 15
  Partial Thromboplastin Time, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Partial Thromboplastin Time, changes to normal or no changes: number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 2 | 15 | 3 | 1 | 5 | 4 | 2 | 15
  Partial Thromboplastin Time, changes to normal or no changes | 1 | 0 | 1 | 0 | 4 | 1 | 8 | 1 | 0 | 4 | 1 | 1 | 7
  Partial Thromboplastin Time, increases to high: number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 2 | 15 | 3 | 1 | 5 | 4 | 2 | 15
  Partial Thromboplastin Time, increases to high | 0 | 1 | 0 | 1 | 3 | 1 | 6 | 2 | 0 | 1 | 3 | 1 | 7
  Prothrombin Intl. Normalized Ratio, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin Intl. Normalized Ratio, changes to normal or no changes | 1 | 1 | 0 | 0 | 4 | 2 | 8 | 1 | 0 | 2 | 2 | 2 | 5
  Prothrombin Intl. Normalized Ratio, increases to high | 0 | 0 | 1 | 1 | 3 | 1 | 10 | 2 | 1 | 5 | 4 | 1 | 10
  Prothrombin Time, decreases to low: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 3 | 16 | 3 | 1 | 6 | 5 | 3 | 15
  Prothrombin Time, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin Time, changes to normal or no changes: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 3 | 16 | 3 | 1 | 6 | 5 | 3 | 15
  Prothrombin Time, changes to normal or no changes | 1 | 1 | 0 | 1 | 3 | 3 | 9 | 1 | 0 | 4 | 3 | 3 | 7
  Prothrombin Time, increases to high: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 3 | 16 | 3 | 1 | 6 | 5 | 3 | 15
  Prothrombin Time, increases to high | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 2 | 1 | 2 | 2 | 0 | 8

8. Primary Outcome: Part 1: Number of Participants With Worst Case Change From Baseline in Urinalysis Parameters
Description: Urine samples were collected for evaluation of urinalysis parameters. The summaries of worst-case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with no change or change to negative and change to positive have been presented.
Time Frame: Baseline (Day 1) and up to 30 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
Participants
  Occult Blood, No Change or Change to Negative | 0 | 1 | 0 | 1 | 5 | 2 | 12 | 2 | 1 | 4 | 4 | 1 | 10
  Occult Blood, Change to Positive | 1 | 0 | 1 | 0 | 2 | 1 | 7 | 1 | 0 | 3 | 2 | 2 | 5
  Protein, No Change or Change to Negative | 1 | 1 | 1 | 1 | 4 | 2 | 11 | 1 | 1 | 2 | 4 | 1 | 10
  Protein, Change to Positive | 0 | 0 | 0 | 0 | 3 | 1 | 8 | 2 | 0 | 5 | 2 | 2 | 5
  Ketones, No Change or Change to Negative | 1 | 1 | 1 | 1 | 5 | 2 | 11 | 2 | 0 | 3 | 3 | 3 | 8
  Ketones, Change to Positive | 0 | 0 | 0 | 0 | 2 | 1 | 8 | 1 | 1 | 4 | 3 | 0 | 7
  Glucose, No Change or Change to Negative | 1 | 1 | 1 | 1 | 7 | 3 | 18 | 3 | 1 | 7 | 5 | 3 | 11
  Glucose, Change to Positive | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4

9. Primary Outcome: Part 1: Changes From Baseline in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected from participants to assess urine pH levels.
Time Frame: Baseline (Day 1) and up to week 132
Population: All treated population. Only those participants with data available at specified timepoint have been analyzed.
Measure: Mean (Standard Deviation); unit: Potential of Hydrogen (pH)
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 3 | 18 | 3 | 1 | 7 | 6 | 3 | 15
Potential of Hydrogen (pH)
  Baseline | 5.00 (NA) — SD could not be calculated for single participant. | 5.50 (NA) — SD could not be calculated for single participant. | 7.00 (NA) — SD could not be calculated for single participant. | 6.50 (NA) — SD could not be calculated for single participant. | 6.00 (0.886) | 6.17 (0.289) | 6.11 (0.698) | 5.67 (0.764) | 6.50 (NA) — SD could not be calculated for single participant. | 5.79 (1.075) | 5.75 (0.524) | 6.17 (0.764) | 5.63 (0.834)
  CFB to Day 8: number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 2 | 18 | 3 | 1 | 7 | 6 | 3 | 15
  CFB to Day 8 | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. | -1.00 (NA) — SD could not be calculated for single participant. | 0.50 (NA) — SD could not be calculated for single participant. | 0.17 (0.516) | -0.25 (0.354) | -0.28 (0.548) | 0.83 (0.764) | 0.50 (NA) — SD could not be calculated for single participant. | -0.07 (1.239) | 0.08 (0.492) | 0.33 (1.258) | -0.03 (0.516)
  CFB to Day 15: number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 3 | 17 | 3 | 1 | 7 | 5 | 1 | 15
  CFB to Day 15 | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. | -1.00 (NA) — SD could not be calculated for single participant. | 0.50 (NA) — SD could not be calculated for single participant. | 0.21 (0.488) | -0.17 (0.289) | -0.24 (0.731) | 0.00 (1.000) | 0.00 (NA) — SD could not be calculated for single participant. | -0.29 (0.859) | 0.10 (0.548) | 1.00 (NA) — SD could not be calculated for single participant. | 0.03 (0.719)
  CFB to Week 4 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 2 | 15 | 3 | 1 | 7 | 5 | 0 | 15
  CFB to Week 4 Day 1 | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. | 0.50 (NA) — SD could not be calculated for single participant. | -0.20 (0.447) | -0.75 (0.354) | -0.13 (0.611) | 0.67 (1.041) | -0.50 (NA) — SD could not be calculated for single participant. | -0.21 (0.488) | 0.10 (0.548) |  | -0.10 (0.849)
  CFB to Week 6 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 2 | 15 | 2 | 1 | 7 | 6 | 2 | 12
  CFB to Week 6 Day 1 | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. | 0.50 (NA) — SD could not be calculated for single participant. | -0.17 (0.577) | 0.00 (0.000) | -0.43 (0.799) | 0.25 (1.061) | -0.50 (NA) — SD could not be calculated for single participant. | -0.29 (1.035) | -0.08 (0.492) | 0.00 (0.707) | -0.04 (0.865)
  CFB to Week 8: number analyzed (Participants) | 1 | 1 | 0 | 1 | 3 | 2 | 13 | 2 | 0 | 4 | 5 | 2 | 9
  CFB to Week 8 | 0.00 (NA) — SD could not be calculated for single participant. | -0.50 (NA) — SD could not be calculated for single participant. |  | 0.50 (NA) — SD could not be calculated for single participant. | -1.17 (1.155) | -0.75 (0.354) | -0.19 (0.630) | 1.00 (0.707) |  | 0.75 (0.645) | -0.20 (0.274) | 0.00 (0.000) | 0.44 (0.682)
  CFB to Week 12: number analyzed (Participants) | 1 | 0 | 0 | 0 | 3 | 1 | 9 | 2 | 0 | 4 | 1 | 2 | 6
  CFB to Week 12 | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  | 0.00 (0.500) | -0.50 (NA) — SD could not be calculated for single participant. | -0.11 (0.546) | 1.00 (1.414) |  | 0.38 (0.629) | 0.00 (NA) — SD could not be calculated for single participant. | -0.25 (1.061) | 0.08 (1.021)
  CFB to Week 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 7 | 2 | 0 | 3 | 1 | 2 | 4
  CFB to Week 16 |  |  |  |  | -0.25 (1.061) | 0.00 (NA) — SD could not be calculated for single participant. | 0.14 (0.690) | 0.50 (1.414) |  | 0.33 (0.289) | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.000) | -0.13 (0.250)
  CFB to Week 20: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 2 | 0 | 3 | 1 | 2 | 4
  CFB to Week 20 |  |  |  |  | -0.75 (0.354) |  | 0.00 (0.548) | -0.50 (0.000) |  | 0.00 (0.000) | 0.00 (NA) — SD could not be calculated for single participant. | 0.50 (0.707) | -0.13 (0.854)
  CFB to Week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 2 | 0 | 2 | 1 | 2 | 5
  CFB to Week 24 |  |  |  |  | -0.75 (1.768) |  | 0.10 (0.418) | 0.75 (1.768) |  | 1.00 (1.414) | 0.00 (NA) — SD could not be calculated for single participant. | 0.50 (0.707) | -0.60 (0.418)
  CFB to Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 2 | 0 | 2 | 0 | 1 | 5
  CFB to Week 28 |  |  |  |  | -1.25 (1.061) |  | -0.13 (0.479) | -0.25 (0.354) |  | 1.50 (0.707) |  | -0.50 (NA) — SD could not be calculated for single participant. | -0.40 (0.418)
  CFB to Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 1 | 0 | 2 | 0 | 2 | 5
  CFB to Week 32 |  |  |  |  | -1.00 (0.707) |  | 0.00 (0.408) | 0.00 (NA) — SD could not be calculated for single participant. |  | 0.25 (0.354) |  | 0.75 (0.354) | 0.10 (1.194)
  CFB to Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 0 | 2 | 0 | 2 | 4
  CFB to Week 36 |  |  |  |  | -1.00 (0.707) |  | 0.00 (0.000) | 0.00 (NA) — SD could not be calculated for single participant. |  | 0.50 (0.000) |  | 0.00 (0.000) | -0.63 (0.479)
  CFB to Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 2 | 0 | 2 | 5
  CFB to Week 40 |  |  |  |  | -1.50 (1.414) |  | -0.17 (0.289) |  |  | 1.00 (1.414) |  | 0.50 (0.707) | -0.20 (0.758)
  CFB to Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 2 | 0 | 1 | 4
  CFB to Week 44 |  |  |  |  | 0.25 (0.354) |  | 0.00 (0.000) |  |  | 0.25 (0.354) |  | 1.50 (NA) — SD could not be calculated for single participant. | -0.13 (0.854)
  CFB to Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 2 | 0 | 1 | 5
  CFB to Week 48 |  |  |  |  | 0.75 (0.354) |  | -0.17 (0.289) |  |  | 0.50 (0.000) |  | 1.00 (NA) — SD could not be calculated for single participant. | -0.50 (0.707)
  CFB to Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 5
  CFB to Week 52 |  |  |  |  | -0.50 (0.707) |  | 0.50 (0.500) |  |  | 0.50 (NA) — SD could not be calculated for single participant. |  | 1.00 (NA) — SD could not be calculated for single participant. | -0.30 (0.274)
  CFB to Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3
  CFB to Week 56 |  |  |  |  |  |  | 0.00 (0.000) |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  | 1.00 (NA) — SD could not be calculated for single participant. | -0.83 (0.289)
  CFB to Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3
  CFB to Week 60 |  |  |  |  |  |  | -0.25 (0.354) |  |  | 0.50 (NA) — SD could not be calculated for single participant. |  | -0.50 (NA) — SD could not be calculated for single participant. | -1.00 (0.500)
  CFB to Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
  CFB to Week 64 |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  | -0.50 (NA) — SD could not be calculated for single participant. | -0.33 (0.764)
  CFB to Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 4
  CFB to Week 68 |  |  |  |  |  |  | -0.25 (0.354) |  |  | 1.50 (NA) — SD could not be calculated for single participant. |  | 0.00 (NA) — SD could not be calculated for single participant. | -0.25 (0.866)
  CFB to Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3
  CFB to Week 72 |  |  |  |  |  |  | -0.25 (0.354) |  |  | 0.50 (NA) — SD could not be calculated for single participant. |  | 0.50 (NA) — SD could not be calculated for single participant. | -0.33 (0.764)
  CFB to Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  CFB to Week 76 |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.50 (NA) — SD could not be calculated for single participant. | -0.75 (0.354)
  CFB to Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  CFB to Week 80 |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  | 1.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.866)
  CFB to Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  CFB to Week 84 |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  | 1.00 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 88: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  CFB to Week 88 |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  | 1.00 (NA) — SD could not be calculated for single participant. | -0.25 (1.061)
  CFB to Week 92: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  CFB to Week 92 |  |  |  |  |  |  | -1.00 (NA) — SD could not be calculated for single participant. |  |  |  |  | 1.00 (NA) — SD could not be calculated for single participant. | -0.75 (0.354)
  CFB to Week 96: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  CFB to Week 96 |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  | 1.00 (NA) — SD could not be calculated for single participant. | -0.33 (0.289)
  CFB to Week 100: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  CFB to Week 100 |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  | 1.00 (NA) — SD could not be calculated for single participant. | -0.25 (0.354)
  CFB to Week 104: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  CFB to Week 104 |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  | 1.00 (NA) — SD could not be calculated for single participant. | -0.83 (0.289)
  CFB to Week 108: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  CFB to Week 108 |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. | -1.00 (0.000)
  CFB to Week 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  CFB to Week 112 |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  | 1.00 (NA) — SD could not be calculated for single participant. | -0.50 (0.866)
  CFB to Week 116: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  CFB to Week 116 |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  | -0.75 (0.354)
  CFB to Week 120: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  CFB to Week 120 |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  | -0.33 (0.289)
  CFB to Week 124: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  CFB to Week 124 |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  | -0.50
  CFB to Week 128: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  CFB to Week 128 |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |  | -0.33 (0.764)
  CFB to Week 132: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 132 |  |  |  |  |  |  | 0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |

10. Primary Outcome: Part 1: Changes From Baseline in Urine Specific Gravity
Description: Urine samples were collected from participants to assess urine specific gravity.
Time Frame: Baseline (Day 1) and up to week 132
Population: All treated population. Only those participants with data available at specified timepoint have been analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 3 | 18 | 3 | 1 | 7 | 6 | 3 | 15
Ratio
  Baseline | 1.02 (NA) — SD could not be calculated for single participant. | 1.03 (NA) — SD could not be calculated for single participant. | 1.01 (NA) — SD could not be calculated for single participant. | 1.02 (NA) — SD could not be calculated for single participant. | 1.02 (0.008) | 1.02 (0.006) | 1.02 (0.007) | 1.02 (0.004) | 1.01 (NA) — SD could not be calculated for single participant. | 1.02 (0.006) | 1.03 (0.008) | 1.02 (0.008) | 1.02 (0.007)
  CFB to Day 8: number analyzed (Participants) | 1 | 1 | 1 | 1 | 6 | 2 | 18 | 3 | 1 | 7 | 6 | 3 | 15
  CFB to Day 8 | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. | 0.01 (NA) — SD could not be calculated for single participant. | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.010) | 0.00 (0.004) | 0.00 (0.007) | 0.00 (0.010) | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.008) | 0.00 (0.006) | 0.00 (0.009) | 0.00 (0.008)
  CFB to Day 15: number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 3 | 17 | 3 | 1 | 7 | 5 | 1 | 15
  CFB to Day 15 | -0.01 (NA) — SD could not be calculated for single participant. | -0.01 (NA) — SD could not be calculated for single participant. | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.010) | -0.01 (0.005) | 0.00 (0.007) | 0.00 (0.005) | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.010) | 0.00 (0.004) | 0.00 | 0.00 (0.008)
  CFB to Week 4 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 5 | 2 | 15 | 3 | 1 | 7 | 5 | 0 | 15
  CFB to Week 4 Day 1 | -0.01 (NA) — SD could not be calculated for single participant. | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.007) | 0.00 (0.004) | 0.00 (0.008) | 0.00 (0.002) | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.007) | 0.00 (0.007) |  | 0.00 (0.007)
  CFB to Week 6 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 2 | 15 | 2 | 1 | 7 | 6 | 2 | 12
  CFB to Week 6 Day 1 | -0.01 (NA) — SD could not be calculated for single participant. | -0.01 (NA) — SD could not be calculated for single participant. | 0.01 (NA) — SD could not be calculated for single participant. | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.008) | -0.01 (0.004) | 0.00 (0.010) | 0.00 (0.006) | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.012) | 0.00 (0.004) | -0.01 (0.007) | 0.00 (0.006)
  CFB to Week 8: number analyzed (Participants) | 1 | 1 | 0 | 1 | 3 | 2 | 13 | 2 | 0 | 4 | 5 | 2 | 9
  CFB to Week 8 | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. |  | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.008) | -0.01 (0.004) | 0.00 (0.008) | 0.00 (0.006) |  | 0.00 (0.006) | 0.00 (0.004) | -0.01 (0.007) | 0.00 (0.007)
  CFB to Week 12: number analyzed (Participants) | 1 | 0 | 0 | 0 | 3 | 1 | 9 | 2 | 0 | 4 | 1 | 2 | 6
  CFB to Week 12 | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  | 0.00 (0.005) | -0.01 | 0.00 (0.008) | -0.01 (0.008) |  | 0.00 (0.010) | -0.01 (NA) — SD could not be calculated for single participant. | -0.01 (0.004) | 0.00 (0.006)
  CFB to Week 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 7 | 2 | 0 | 3 | 1 | 2 | 4
  CFB to Week 16 |  |  |  |  | 0.00 (0.011) | -0.02 (NA) — SD could not be calculated for single participant. | 0.00 (0.006) | -0.01 (0.004) |  | -0.01 (0.008) | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.004) | 0.00 (0.004)
  CFB to Week 20: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 2 | 0 | 3 | 1 | 2 | 4
  CFB to Week 20 |  |  |  |  | 0.00 (0.004) |  | 0.00 (0.008) | 0.00 (0.002) |  | 0.00 (0.007) | 0.00 (NA) — SD could not be calculated for single participant. | -0.01 (0.004) | 0.00 (0.003)
  CFB to Week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 2 | 0 | 2 | 1 | 2 | 5
  CFB to Week 24 |  |  |  |  | 0.00 (0.011) |  | 0.00 (0.004) | 0.00 (0.004) |  | 0.00 (0.006) | 0.00 (NA) — SD could not be calculated for single participant. | -0.01 (0.000) | 0.00 (0.002)
  CFB to Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 2 | 0 | 2 | 0 | 1 | 5
  CFB to Week 28 |  |  |  |  | 0.00 (0.011) |  | 0.00 (0.012) | 0.00 (0.004) |  | 0.00 (0.015) |  | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.006)
  CFB to Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 1 | 0 | 2 | 0 | 2 | 5
  CFB to Week 32 |  |  |  |  | 0.00 (0.004) |  | 0.00 (0.007) | 0.01 (NA) — SD could not be calculated for single participant. |  | 0.00 (0.014) |  | 0.00 (0.004) | 0.00 (0.003)
  CFB to Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 0 | 2 | 0 | 2 | 4
  CFB to Week 36 |  |  |  |  | -0.01 (0.014) |  | 0.01 (0.013) | 0.01 (NA) — SD could not be calculated for single participant. |  | 0.00 (0.008) |  | 0.01 (0.011) | 0.00 (0.002)
  CFB to Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 2 | 0 | 2 | 5
  CFB to Week 40 |  |  |  |  | 0.00 (0.014) |  | 0.00 (0.012) |  |  | 0.00 (0.015) |  | -0.01 (0.000) | 0.00 (0.003)
  CFB to Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 2 | 0 | 1 | 4
  CFB to Week 44 |  |  |  |  | 0.00 (0.014) |  | 0.00 (0.008) |  |  | 0.00 (0.010) |  | -0.01 | 0.00 (0.004)
  CFB to Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 2 | 0 | 1 | 5
  CFB to Week 48 |  |  |  |  | -0.01 (0.014) |  | 0.00 (0.006) |  |  | 0.00 (0.010) |  | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.005)
  CFB to Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 5
  CFB to Week 52 |  |  |  |  | 0.00 (0.018) |  | 0.00 (0.009) |  |  | 0.01 (NA) — SD could not be calculated for single participant. |  | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.004)
  CFB to Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3
  CFB to Week 56 |  |  |  |  |  |  | -0.01 (0.004) |  |  | 0.01 (NA) — SD could not be calculated for single participant. |  | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.005)
  CFB to Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3
  CFB to Week 60 |  |  |  |  |  |  | -0.01 (0.004) |  |  | 0.01 (NA) — SD could not be calculated for single participant. |  | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.006)
  CFB to Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
  CFB to Week 64 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  | 0.01 (NA) — SD could not be calculated for single participant. |  | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.007)
  CFB to Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 4
  CFB to Week 68 |  |  |  |  |  |  | -0.01 (0.000) |  |  | 0.01 (NA) — SD could not be calculated for single participant. |  | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.003)
  CFB to Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 3
  CFB to Week 72 |  |  |  |  |  |  | 0.00 (0.007) |  |  | 0.01 (NA) — SD could not be calculated for single participant. |  | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.002)
  CFB to Week 76: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  CFB to Week 76 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.004)
  CFB to Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  CFB to Week 80 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.006)
  CFB to Week 84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  CFB to Week 84 |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 88: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  CFB to Week 88 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.003)
  CFB to Week 92: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  CFB to Week 92 |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.006)
  CFB to Week 96: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  CFB to Week 96 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.003)
  CFB to Week 100: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  CFB to Week 100 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.001)
  CFB to Week 104: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  CFB to Week 104 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.01 (NA) — SD could not be calculated for single participant. | -0.01 (0.008)
  CFB to Week 108: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  CFB to Week 108 |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.004)
  CFB to Week 112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  CFB to Week 112 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.007)
  CFB to Week 116: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  CFB to Week 116 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  | 0.00 (0.004)
  CFB to Week 120: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  CFB to Week 120 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  | 0.01 (0.008)
  CFB to Week 124: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  CFB to Week 124 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  | 0.01 (NA) — SD could not be calculated for single participant.
  CFB to Week 128: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  CFB to Week 128 |  |  |  |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  | 0.01 (0.008)
  CFB to Week 132: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 132 |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |

11. Primary Outcome: Part 1: Number of Participants With Maximum Grade Worst Case Increase Post-baseline Relative to Baseline in Vital Signs
Description: The abnormal vital sign ranges are: Heart Rate:- Low (<60 beats per minute (bpm)), Normal (>=60 bpm to <=100 bpm), High (>100 bpm); Temperature:- Low (<=35 degree Celsius (°C)), Normal (>35 °C and <38 °C), High (>=38 °C); Systolic Blood Pressure:- Low (<90 millimeter of mercury (mmHg)), Normal (>=90 mmHg to <120 mmHg), High (>=120 mmHg); Diastolic Blood Pressure:- Low (<60 mmHg), Normal (>=60 mmHg to <80 mmHg), High (>=80 mmHg). Participants were counted in the worst-case category and their value changes to (low, normal or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Baseline (Day 1) and up to 30 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
Participants
  Heart Rate, changes to low | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2
  Heart Rate, changes to normal or no changes | 1 | 1 | 1 | 0 | 5 | 3 | 12 | 3 | 1 | 3 | 6 | 2 | 10
  Heart Rate, changes to high | 0 | 0 | 0 | 1 | 1 | 0 | 6 | 0 | 0 | 3 | 0 | 1 | 3
  Temperature, changes to low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature, changes to normal or no changes | 1 | 1 | 1 | 1 | 6 | 3 | 17 | 3 | 1 | 6 | 6 | 3 | 15
  Temperature, changes to high | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  Systolic Blood Pressure, changes to low | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 2
  Systolic Blood Pressure, changes to normal or no changes | 0 | 1 | 1 | 1 | 5 | 2 | 9 | 1 | 1 | 5 | 5 | 1 | 11
  Systolic Blood Pressure, changes to high | 1 | 0 | 0 | 0 | 2 | 1 | 7 | 1 | 0 | 1 | 1 | 2 | 2
  Diastolic Blood Pressure, changes to low | 0 | 0 | 0 | 0 | 1 | 2 | 6 | 1 | 0 | 0 | 0 | 1 | 3
  Diastolic Blood Pressure, changes to normal or no changes | 1 | 0 | 1 | 0 | 4 | 1 | 7 | 0 | 1 | 7 | 4 | 1 | 8
  Diastolic Blood Pressure, changes to high | 0 | 1 | 0 | 1 | 2 | 1 | 8 | 3 | 0 | 0 | 2 | 1 | 5

12. Primary Outcome: Part 3: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or was a congenital anomaly/birth defect, other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function. SAEs are subset of AEs. A summary of number of participants with any AEs and SAEs is presented. AEs were coded using the MedDRA dictionary.
Time Frame: Up to 10 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 10
Participants
  Any AEs | 9
  Any SAEs | 5

13. Primary Outcome: Part 3: Number of Participants Withdrawn Due to AEs
Description: The data for number of participants withdrawn due to AEs have been presented.
Time Frame: Up to 10 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 10
Participants | 1

14. Primary Outcome: Part 3: Number of Participants With Dose Modifications of GSK3326595 and Pembrolizumab
Description: The number of participants who experienced any dose modifications (interruptions and reductions) of GSK3326595 and pembrolizumab have been presented.
Time Frame: Up to 10 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 10
Participants
  Dose interruptions of GSK3326595 | 1
  Dose reductions of GSK3326595 | 0
  Dose Interruptions of Pembrolizumab | 1
  Dose reductions of Pembrolizumab | 0

15. Primary Outcome: Part 3: Number of Participants With Worst Case Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for evaluation of clinical chemistry parameters. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with decreases to low, changes to normal or no changes from Baseline, and increases to high values have been presented.
Time Frame: Baseline (Day 1) and up to 10 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 9
Participants
  Alanine Aminotransferase, decreases to low | 2
  Alanine Aminotransferase, changes to normal or no changes | 3
  Alanine Aminotransferase, increases to high | 4
  Albumin, decreases to low | 3
  Albumin, changes to normal or no changes | 6
  Albumin, increases to high | 0
  Alkaline Phosphatase, decreases to low | 0
  Alkaline Phosphatase, changes to normal or no changes | 8
  Alkaline Phosphatase, increases to high | 1
  Amylase, decreases to low | 2
  Amylase, changes to normal or no changes | 6
  Amylase, increases to high | 1
  Aspartate Aminotransferase, decreases to low | 0
  Aspartate Aminotransferase, changes to normal or no changes | 6
  Aspartate Aminotransferase, increases to high | 3
  Bilirubin, decreases to low | 0
  Bilirubin, changes to normal or no changes | 7
  Bilirubin, increases to high | 2
  Calcium, decreases to low | 7
  Calcium, changes to normal or no changes | 2
  Calcium, increases to high | 0
  Creatinine, decreases to low | 0
  Creatinine, changes to normal or no changes | 8
  Creatinine, increases to high | 1
  Direct Bilirubin, decreases to low | 0
  Direct Bilirubin, changes to normal or no changes | 6
  Direct Bilirubin, increases to high | 3
  Glucose, decreases to low | 0
  Glucose, changes to normal or no changes | 7
  Glucose, increases to high | 2
  Lipase, decreases to low | 2
  Lipase, changes to normal or no changes | 6
  Lipase, increases to high | 1
  Potassium, decreases to low | 4
  Potassium, changes to normal or no changes | 4
  Potassium, increases to high | 1
  Protein, decreases to low | 5
  Protein, changes to normal or no changes | 3
  Protein, increases to high | 1
  Sodium, decreases to low | 2
  Sodium, changes to normal or no changes | 6
  Sodium, increases to high | 1
  Urea Nitrogen, decreases to low: number analyzed (Participants) | 5
  Urea Nitrogen, decreases to low | 0
  Urea Nitrogen, changes to normal or no changes: number analyzed (Participants) | 5
  Urea Nitrogen, changes to normal or no changes | 4
  Urea Nitrogen, increases to high: number analyzed (Participants) | 5
  Urea Nitrogen, increases to high | 1

16. Primary Outcome: Part 3: Number of Participants With Worst Case Change From Baseline in Hematology Parameters
Description: Blood samples were collected for evaluation of hematology parameters. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with decreases to low, changes to normal or no changes from Baseline, and increases to high values have been presented.
Time Frame: Baseline (Day 1) and up to 10 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 9
Participants
  Basophils, decreases to low | 0
  Basophils, changes to normal or no changes | 9
  Basophils, increases to high | 0
  Eosinophils, decreases to low | 0
  Eosinophils, changes to normal or no changes | 8
  Eosinophils, increases to high | 1
  Mean Corpuscular Hemoglobin, decreases to low | 1
  Mean Corpuscular Hemoglobin, changes to normal or no changes | 8
  Mean Corpuscular Hemoglobin, increases to high | 0
  Mean Corpuscular Volume, decreases to low | 1
  Mean Corpuscular Volume, changes to normal or no changes | 7
  Mean Corpuscular Volume, increases to high | 1
  Erythrocytes, decreases to low | 1
  Erythrocytes, changes to normal or no changes | 8
  Erythrocytes, increases to high | 0
  Hematocrit, decreases to low | 0
  Hematocrit, changes to normal or no changes | 9
  Hematocrit, increases to high | 0
  Hemoglobin, decreases to low | 2
  Hemoglobin, changes to normal or no changes | 7
  Hemoglobin, increases to high | 0
  Leukocytes, decreases to low | 3
  Leukocytes, changes to normal or no changes | 5
  Leukocytes, increases to high | 1
  Lymphocytes, decreases to low | 5
  Lymphocytes, changes to normal or no changes | 4
  Lymphocytes, increases to high | 0
  Monocytes, decreases to low | 0
  Monocytes, changes to normal or no changes | 8
  Monocytes, increases to high | 1
  Neutrophils, decreases to low | 1
  Neutrophils, changes to normal or no changes | 7
  Neutrophils, increases to high | 1
  Platelets, decreases to low | 1
  Platelets, changes to normal or no changes | 6
  Platelets, increases to high | 2
  Reticulocytes, decreases to low: number analyzed (Participants) | 8
  Reticulocytes, decreases to low | 0
  Reticulocytes, changes to normal or no changes: number analyzed (Participants) | 8
  Reticulocytes, changes to normal or no changes | 5
  Reticulocytes, increases to high: number analyzed (Participants) | 8
  Reticulocytes, increases to high | 3

17. Primary Outcome: Part 3: Number of Participants With Worst Case Change From Baseline in Coagulation Parameters
Description: Blood samples were collected for evaluation of coagulation parameters. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with 'decreases to low', 'changes to normal' or 'no changes from Baseline', and 'increases to high' values have been presented.
Time Frame: Baseline (Day 1) and up to 10 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 9
Participants
  Partial Thromboplastin Time, decreases to low | 1
  Partial Thromboplastin Time, changes to normal or no changes | 5
  Partial Thromboplastin Time, increases to high | 3
  Prothrombin Intl. Normalized Ratio, decreases to low | 1
  Prothrombin Intl. Normalized Ratio, changes to normal or no changes | 6
  Prothrombin Intl. Normalized Ratio, increases to high | 2
  Prothrombin Time, decreases to low | 1
  Prothrombin Time, changes to normal or no changes | 4
  Prothrombin Time, increases to high | 4

18. Primary Outcome: Part 3: Number of Participants With Worst Case Change From Baseline in Urinalysis Parameters
Description: Urine samples were collected for evaluation of urinalysis parameters. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with no change or change to negative and change to positive values have been presented.
Time Frame: Baseline (Day 1) and up to 10 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 10
Participants
  Occult Blood, No Change or Change to Negative | 7
  Occult Blood, Change to Positive | 3
  Protein, No Change or Change to Negative | 8
  Protein, Change to Positive | 2
  Ketones, No Change or Change to Negative | 7
  Ketones, Change to Positive | 3
  Glucose, No Change or Change to Negative | 10
  Glucose, Change to Positive | 0

19. Primary Outcome: Part 3: Changes From Baseline in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected from participants to assess urine pH levels.
Time Frame: Baseline (Day 1) and up to Week 42
Population: All treated population. Only those participants with data available at specified timepoint have been analyzed.
Measure: Mean (Standard Deviation); unit: Potential of Hydrogen (pH)
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 10
Potential of Hydrogen (pH)
  Baseline | 5.60 (0.937)
  CFB to Day 1: number analyzed (Participants) | 1
  CFB to Day 1 | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Day 8: number analyzed (Participants) | 8
  CFB to Day 8 | 0.38 (0.582)
  CFB to Day 15: number analyzed (Participants) | 9
  CFB to Day 15 | 0.33 (0.750)
  CFB to Week 4 Day 1: number analyzed (Participants) | 9
  CFB to Week 4 Day 1 | 0.33 (0.500)
  Week 6 Day 1: number analyzed (Participants) | 8
  Week 6 Day 1 | 0.31 (0.704)
  CFB to Week 8: number analyzed (Participants) | 2
  CFB to Week 8 | 0.25 (0.354)
  CFB to Week 9: number analyzed (Participants) | 3
  CFB to Week 9 | 0.33 (0.577)
  CFB to Week 12: number analyzed (Participants) | 3
  CFB to Week 12 | 0.83 (0.764)
  CFB to Week 15: number analyzed (Participants) | 3
  CFB to Week 15 | 0.67 (0.289)
  CFB to Week 18: number analyzed (Participants) | 3
  CFB to Week 18 | 0.50 (0.500)
  CFB to Week 21: number analyzed (Participants) | 3
  CFB to Week 21 | 0.50 (0.500)
  CFB to Week 24: number analyzed (Participants) | 2
  CFB to Week 24 | 0.25 (0.354)
  CFB to Week 27: number analyzed (Participants) | 2
  CFB to Week 27 | 0.25 (0.354)
  CFB to Week 30: number analyzed (Participants) | 1
  CFB to Week 30 | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 33: number analyzed (Participants) | 1
  CFB to Week 33 | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 36: number analyzed (Participants) | 1
  CFB to Week 36 | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 39: number analyzed (Participants) | 1
  CFB to Week 39 | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 42: number analyzed (Participants) | 1
  CFB to Week 42 | 0.00 (NA) — SD could not be calculated for single participant.

20. Primary Outcome: Part 3: Changes From Baseline in Urine Specific Gravity
Description: Urine samples were collected from participants to assess urine specific gravity.
Time Frame: Baseline (Day 1) and up to Week 42
Population: All treated population. Only those participants with data available at specified timepoint have been analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 10
Ratio
  Baseline | 1.02 (0.008)
  CFB to Day 1: number analyzed (Participants) | 1
  CFB to Day 1 | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Day 8: number analyzed (Participants) | 8
  CFB to Day 8 | -0.01 (0.009)
  CFB to Day 15: number analyzed (Participants) | 9
  CFB to Day 15 | 0.00 (0.006)
  CFB to Week 4 Day 1: number analyzed (Participants) | 9
  CFB to Week 4 Day 1 | -0.01 (0.008)
  CFB to Week 6 Day 1: number analyzed (Participants) | 8
  CFB to Week 6 Day 1 | 0.00 (0.007)
  CFB to Week 8: number analyzed (Participants) | 2
  CFB to Week 8 | 0.00 (0.001)
  CFB to Week 9: number analyzed (Participants) | 3
  CFB to Week 9 | -0.01 (0.003)
  CFB to Week 12: number analyzed (Participants) | 3
  CFB to Week 12 | -0.01 (0.006)
  CFB to Week 15: number analyzed (Participants) | 3
  CFB to Week 15 | 0.00 (0.008)
  CFB to Week 18: number analyzed (Participants) | 3
  CFB to Week 18 | -0.01 (0.007)
  CFB to Week 21: number analyzed (Participants) | 3
  CFB to Week 21 | 0.00 (0.009)
  CFB to Week 24: number analyzed (Participants) | 2
  CFB to Week 24 | -0.01 (0.001)
  CFB to Week 27: number analyzed (Participants) | 2
  CFB to Week 27 | 0.00 (0.016)
  CFB to Week 30: number analyzed (Participants) | 1
  CFB to Week 30 | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 33: number analyzed (Participants) | 1
  CFB to Week 33 | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 36: number analyzed (Participants) | 1
  CFB to Week 36 | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 39: number analyzed (Participants) | 1
  CFB to Week 39 | 0.01 (NA) — SD could not be calculated for single participant.
  CFB to Week 42: number analyzed (Participants) | 1
  CFB to Week 42 | 0.01 (NA) — SD could not be calculated for single participant.

21. Primary Outcome: Part 3: Number of Participants With Maximum Worst-case Increase Post-baseline Relative to Baseline in Vital Signs
Description: The abnormal vital sign ranges are: Heart Rate:- Low [<60 bpm], Normal (>=60 bpm to <=100 bpm), High (>100 bpm); Temperature:- Low (<=35 C), Normal (>35 C and <38 C), High (>=38 C); Systolic Blood Pressure:- Low (<90 mmHg), Normal (>=90 mmHg to <120 mmHg), High (>=120 mmHg); Diastolic Blood Pressure:- Low (<60 mmHg), Normal (>=60 mmHg to <80 mmHg), High (>=80 mmHg). Participants were counted in the maximum worst case increase category that their value changes to (low, normal or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Baseline (Day 1) and up to 10 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 9
Participants
  Heart Rate, changes to low | 0
  Heart Rate, changes to normal or no changes | 6
  Heart Rate, changes to high | 3
  Temperature, changes to low | 0
  Temperature, changes to normal or no changes | 9
  Temperature, changes to high | 0
  Systolic Blood Pressure, changes to low | 0
  Systolic Blood Pressure, changes to normal or no changes | 5
  Systolic Blood Pressure, changes to high | 4
  Diastolic Blood Pressure, changes to low | 2
  Diastolic Blood Pressure, changes to normal or no changes | 2
  Diastolic Blood Pressure, changes to high | 6

22. Secondary Outcome: Part 2: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or is a congenital anomaly/birth defect, other situations which involved medical or scientific judgment or was associated with liver injury and impaired liver function. SAEs are subset of AEs. AEs were coded using the MedDRA dictionary.
Time Frame: Up to 42 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC)
Number analyzed (Participants) | 22 | 16 | 29 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
Participants
  Any AEs | 22 | 16 | 27 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
  Any SAEs | 13 | 7 | 15 | 10 | 13 | 15 | 5 | 4 | 2 | 4 | 0 | 4 | 0

23. Secondary Outcome: Part 2: Number of Participants Withdrawn Due to AEs
Description: The data for number of participants withdrawn due to AEs have been presented.
Time Frame: Up to 42 months
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC)
Number analyzed (Participants) | 22 | 16 | 29 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
Participants | 4 | 4 | 4 | 3 | 1 | 3 | 2 | 1 | 0 | 1 | 0 | 3 | 1

24. Secondary Outcome: Part 2: Number of Participants With Dose Modifications of GSK3326595
Description: The number of participants who had any dose modifications (interruptions and reductions) of GSK3326595 have been presented.
Time Frame: Up to 42 months
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC)
Number analyzed (Participants) | 22 | 16 | 29 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
Participants
  Dose interruptions | 13 | 12 | 11 | 22 | 20 | 28 | 13 | 4 | 2 | 3 | 2 | 5 | 2
  Dose reductions | 8 | 11 | 11 | 26 | 18 | 27 | 7 | 4 | 2 | 4 | 0 | 6 | 3

25. Secondary Outcome: Part 2: Number of Participants With Worst Case Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for evaluation of clinical chemistry parameters. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with 'decreases to low', 'changes to normal' or 'no changes from Baseline', and 'increases to high' values have been presented. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Baseline (Day 1) and up to 42 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC)
Number analyzed (Participants) | 22 | 16 | 28 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
Participants
  Alanine Aminotransferase, decreases to low | 1 | 1 | 0 | 2 | 1 | 9 | 7 | 0 | 0 | 0 | 0 | 0 | 1
  Alanine Aminotransferase, changes to normal or no changes | 20 | 12 | 24 | 30 | 25 | 23 | 9 | 5 | 2 | 7 | 2 | 10 | 6
  Alanine Aminotransferase, increases to high | 1 | 3 | 4 | 6 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0
  Albumin, decreases to low | 8 | 6 | 6 | 15 | 11 | 19 | 7 | 3 | 0 | 4 | 0 | 3 | 0
  Albumin, changes to normal or no changes | 14 | 10 | 22 | 22 | 17 | 14 | 9 | 3 | 2 | 4 | 2 | 8 | 7
  Albumin, increases to high | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase, changes to normal or no changes | 19 | 10 | 27 | 30 | 24 | 26 | 14 | 3 | 1 | 5 | 2 | 9 | 4
  Alkaline Phosphatase, increases to high | 3 | 6 | 1 | 7 | 4 | 8 | 2 | 2 | 1 | 3 | 0 | 2 | 3
  Amylase, decreases to low | 1 | 1 | 0 | 4 | 4 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Amylase, changes to normal or no changes | 19 | 10 | 25 | 31 | 23 | 28 | 14 | 3 | 2 | 7 | 2 | 10 | 5
  Amylase, increases to high | 2 | 5 | 3 | 2 | 2 | 5 | 1 | 2 | 0 | 1 | 0 | 1 | 0
  Aspartate Aminotransferase, decreases to low | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Aspartate Aminotransferase, changes to normal or no changes | 15 | 12 | 25 | 30 | 22 | 19 | 15 | 4 | 1 | 6 | 1 | 8 | 6
  Aspartate Aminotransferase, increases to high | 7 | 4 | 3 | 7 | 6 | 13 | 0 | 2 | 1 | 2 | 1 | 2 | 1
  Bilirubin, decreases to low | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Bilirubin, changes to normal or no changes | 17 | 11 | 22 | 30 | 25 | 30 | 11 | 5 | 1 | 7 | 2 | 10 | 7
  Bilirubin, increases to high | 5 | 5 | 5 | 7 | 3 | 4 | 4 | 1 | 1 | 0 | 0 | 1 | 0
  Calcium, decreases to low | 6 | 7 | 9 | 8 | 10 | 11 | 3 | 6 | 1 | 5 | 0 | 5 | 3
  Calcium, changes to normal or no changes | 16 | 9 | 19 | 25 | 17 | 23 | 13 | 0 | 1 | 3 | 2 | 5 | 4
  Calcium, increases to high | 0 | 1 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine, decreases to low | 5 | 0 | 3 | 5 | 5 | 6 | 4 | 0 | 0 | 0 | 1 | 1 | 1
  Creatinine, changes to normal or no changes | 15 | 10 | 22 | 24 | 17 | 25 | 12 | 3 | 2 | 6 | 1 | 7 | 5
  Creatinine, increases to high | 2 | 6 | 3 | 8 | 6 | 3 | 1 | 3 | 0 | 2 | 0 | 3 | 1
  Direct Bilirubin, decreases to low: number analyzed (Participants) | 22 | 16 | 28 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 10 | 7
  Direct Bilirubin, decreases to low | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin, changes to normal or no changes: number analyzed (Participants) | 22 | 16 | 28 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 10 | 7
  Direct Bilirubin, changes to normal or no changes | 15 | 7 | 16 | 27 | 23 | 20 | 10 | 4 | 1 | 5 | 0 | 6 | 7
  Direct Bilirubin, increases to high: number analyzed (Participants) | 22 | 16 | 28 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 10 | 7
  Direct Bilirubin, increases to high | 7 | 9 | 12 | 10 | 5 | 14 | 6 | 2 | 1 | 3 | 2 | 4 | 0
  Glucose, decreases to low | 2 | 2 | 0 | 3 | 2 | 4 | 2 | 0 | 0 | 1 | 0 | 0 | 2
  Glucose, changes to normal or no changes | 14 | 10 | 25 | 24 | 13 | 16 | 9 | 3 | 1 | 2 | 2 | 7 | 3
  Glucose, increases to high | 6 | 5 | 3 | 10 | 14 | 15 | 6 | 3 | 1 | 6 | 0 | 4 | 2
  Lipase, decreases to low | 1 | 1 | 1 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1
  Lipase, changes to normal or no changes | 19 | 12 | 21 | 31 | 25 | 26 | 15 | 4 | 2 | 7 | 1 | 11 | 5
  Lipase, increases to high | 2 | 3 | 6 | 5 | 3 | 6 | 0 | 1 | 0 | 1 | 1 | 0 | 1
  Potassium, decreases to low | 3 | 4 | 3 | 5 | 5 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0
  Potassium, changes to normal or no changes | 18 | 11 | 21 | 25 | 19 | 23 | 12 | 2 | 1 | 6 | 1 | 10 | 4
  Potassium, increases to high | 2 | 2 | 4 | 7 | 6 | 10 | 3 | 4 | 0 | 2 | 1 | 0 | 3
  Protein, decreases to low | 8 | 4 | 12 | 7 | 12 | 13 | 7 | 4 | 1 | 5 | 1 | 7 | 3
  Protein, changes to normal or no changes | 13 | 10 | 16 | 28 | 16 | 20 | 9 | 2 | 1 | 3 | 1 | 4 | 4
  Protein, increases to high | 1 | 3 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, decreases to low | 6 | 5 | 1 | 8 | 6 | 6 | 4 | 1 | 0 | 1 | 0 | 3 | 1
  Sodium, changes to normal or no changes | 13 | 9 | 25 | 29 | 22 | 25 | 10 | 4 | 2 | 7 | 2 | 7 | 6
  Sodium, increases to high | 3 | 2 | 2 | 1 | 0 | 4 | 2 | 1 | 0 | 0 | 0 | 1 | 0
  Urea Nitrogen, decreases to low: number analyzed (Participants) | 3 | 10 | 14 | 17 | 14 | 17 | 14 | 2 | 0 | 3 | 0 | 5 | 2
  Urea Nitrogen, decreases to low | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 0 |  | 0 |  | 0 | 0
  Urea Nitrogen, changes to normal or no changes: number analyzed (Participants) | 3 | 10 | 14 | 17 | 14 | 17 | 14 | 2 | 0 | 3 | 0 | 5 | 2
  Urea Nitrogen, changes to normal or no changes | 3 | 5 | 9 | 11 | 7 | 8 | 6 | 0 |  | 3 |  | 2 | 1
  Urea Nitrogen, increases to high: number analyzed (Participants) | 3 | 10 | 14 | 17 | 14 | 17 | 14 | 2 | 0 | 3 | 0 | 5 | 2
  Urea Nitrogen, increases to high | 0 | 5 | 5 | 5 | 6 | 8 | 6 | 2 |  | 0 |  | 3 | 1

26. Secondary Outcome: Part 2: Number of Participants With Worst Case Change From Baseline in Hematology Parameters
Description: Blood samples were collected for evaluation of hematology parameters. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with 'decreases to low', 'changes to normal' or 'no changes from Baseline', and 'increases to high values' have been presented. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Baseline (Day 1) and up to 42 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC)
Number analyzed (Participants) | 22 | 16 | 28 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
Participants
  Basophils, decreases to low: number analyzed (Participants) | 21 | 16 | 25 | 37 | 28 | 34 | 16 | 5 | 2 | 6 | 2 | 8 | 7
  Basophils, decreases to low | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils, changes to normal or no changes: number analyzed (Participants) | 21 | 16 | 25 | 37 | 28 | 34 | 16 | 5 | 2 | 6 | 2 | 8 | 7
  Basophils, changes to normal or no changes | 21 | 16 | 24 | 35 | 26 | 33 | 16 | 5 | 2 | 5 | 2 | 8 | 7
  Basophils, increases to high: number analyzed (Participants) | 21 | 16 | 25 | 37 | 28 | 34 | 16 | 5 | 2 | 6 | 2 | 8 | 7
  Basophils, increases to high | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Eosinophils, decreases to low: number analyzed (Participants) | 21 | 16 | 25 | 37 | 28 | 34 | 16 | 5 | 2 | 6 | 2 | 8 | 7
  Eosinophils, decreases to low | 0 | 0 | 2 | 2 | 2 | 3 | 2 | 1 | 0 | 0 | 0 | 2 | 0
  Eosinophils, changes to normal or no changes: number analyzed (Participants) | 21 | 16 | 25 | 37 | 28 | 34 | 16 | 5 | 2 | 6 | 2 | 8 | 7
  Eosinophils, changes to normal or no changes | 21 | 14 | 23 | 33 | 26 | 29 | 14 | 4 | 2 | 6 | 2 | 5 | 4
  Eosinophils, increases to high: number analyzed (Participants) | 21 | 16 | 25 | 37 | 28 | 34 | 16 | 5 | 2 | 6 | 2 | 8 | 7
  Eosinophils, increases to high | 0 | 2 | 0 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  Mean Corpuscular Hemoglobin, decreases to low: number analyzed (Participants) | 22 | 16 | 28 | 36 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
  Mean Corpuscular Hemoglobin, decreases to low | 3 | 0 | 0 | 5 | 3 | 6 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Hemoglobin, changes to normal or no changes: number analyzed (Participants) | 22 | 16 | 28 | 36 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
  Mean Corpuscular Hemoglobin, changes to normal or no changes | 18 | 16 | 26 | 28 | 25 | 26 | 12 | 5 | 2 | 8 | 2 | 11 | 7
  Mean Corpuscular Hemoglobin, increases to high: number analyzed (Participants) | 22 | 16 | 28 | 36 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
  Mean Corpuscular Hemoglobin, increases to high | 1 | 0 | 2 | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Corpuscular Volume, decreases to low | 1 | 2 | 0 | 5 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  Mean Corpuscular Volume, changes to normal or no changes | 20 | 11 | 28 | 29 | 28 | 29 | 13 | 4 | 2 | 7 | 2 | 9 | 7
  Mean Corpuscular Volume, increases to high | 1 | 3 | 0 | 3 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 2 | 0
  Erythrocytes, decreases to low: number analyzed (Participants) | 22 | 16 | 28 | 36 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
  Erythrocytes, decreases to low | 13 | 7 | 11 | 17 | 12 | 22 | 10 | 2 | 1 | 3 | 2 | 1 | 3
  Erythrocytes, changes to normal or no changes: number analyzed (Participants) | 22 | 16 | 28 | 36 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
  Erythrocytes, changes to normal or no changes | 9 | 9 | 17 | 19 | 16 | 12 | 5 | 3 | 1 | 5 | 0 | 10 | 4
  Erythrocytes, increases to high: number analyzed (Participants) | 22 | 16 | 28 | 36 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
  Erythrocytes, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
  Hematocrit, decreases to low | 11 | 9 | 13 | 18 | 12 | 24 | 10 | 3 | 1 | 6 | 2 | 5 | 4
  Hematocrit, changes to normal or no changes | 11 | 7 | 15 | 19 | 16 | 10 | 6 | 3 | 1 | 2 | 0 | 6 | 3
  Hematocrit, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, decreases to low | 13 | 8 | 13 | 21 | 11 | 22 | 10 | 3 | 1 | 5 | 2 | 5 | 5
  Hemoglobin, changes to normal or no changes | 9 | 8 | 15 | 16 | 17 | 12 | 6 | 3 | 1 | 3 | 0 | 6 | 2
  Hemoglobin, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes, decreases to low | 11 | 4 | 9 | 15 | 16 | 15 | 8 | 2 | 1 | 5 | 1 | 10 | 1
  Leukocytes, changes to normal or no changes | 10 | 8 | 18 | 20 | 9 | 15 | 6 | 3 | 0 | 3 | 1 | 1 | 4
  Leukocytes, increases to high | 3 | 4 | 1 | 2 | 4 | 4 | 4 | 1 | 1 | 1 | 0 | 1 | 2
  Lymphocytes, decreases to low | 8 | 6 | 8 | 8 | 11 | 15 | 7 | 1 | 1 | 1 | 0 | 3 | 3
  Lymphocytes, changes to normal or no changes | 14 | 10 | 20 | 29 | 17 | 19 | 9 | 5 | 0 | 7 | 2 | 8 | 4
  Lymphocytes, increases to high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Monocytes, decreases to low: number analyzed (Participants) | 21 | 16 | 25 | 37 | 28 | 34 | 16 | 5 | 2 | 6 | 2 | 8 | 7
  Monocytes, decreases to low | 5 | 1 | 3 | 5 | 5 | 6 | 1 | 1 | 1 | 2 | 0 | 2 | 0
  Monocytes, changes to normal or no changes: number analyzed (Participants) | 21 | 16 | 25 | 37 | 28 | 34 | 16 | 5 | 2 | 6 | 2 | 8 | 7
  Monocytes, changes to normal or no changes | 14 | 11 | 20 | 28 | 19 | 20 | 9 | 3 | 0 | 3 | 1 | 4 | 6
  Monocytes, increases to high: number analyzed (Participants) | 21 | 16 | 25 | 37 | 28 | 34 | 16 | 5 | 2 | 6 | 2 | 8 | 7
  Monocytes, increases to high | 4 | 5 | 3 | 4 | 5 | 10 | 6 | 1 | 1 | 2 | 1 | 2 | 1
  Neutrophils, decreases to low | 8 | 2 | 6 | 12 | 7 | 8 | 5 | 3 | 2 | 4 | 1 | 7 | 1
  Neutrophils, changes to normal or no changes | 12 | 11 | 19 | 22 | 18 | 22 | 7 | 2 | 0 | 1 | 1 | 2 | 4
  Neutrophils, increases to high | 2 | 3 | 3 | 3 | 3 | 4 | 4 | 2 | 0 | 4 | 0 | 4 | 2
  Platelets, decreases to low | 14 | 13 | 8 | 17 | 20 | 14 | 5 | 3 | 1 | 5 | 1 | 9 | 2
  Platelets, changes to normal or no changes | 6 | 3 | 20 | 18 | 8 | 14 | 10 | 2 | 1 | 3 | 1 | 2 | 4
  Platelets, increases to high | 3 | 3 | 1 | 2 | 1 | 10 | 2 | 1 | 0 | 0 | 0 | 1 | 1
  Reticulocytes, decreases to low: number analyzed (Participants) | 22 | 16 | 28 | 32 | 26 | 34 | 15 | 6 | 2 | 8 | 2 | 11 | 7
  Reticulocytes, decreases to low | 9 | 12 | 8 | 9 | 15 | 19 | 5 | 2 | 1 | 1 | 0 | 5 | 2
  Reticulocytes, changes to normal or no changes: number analyzed (Participants) | 22 | 16 | 28 | 32 | 26 | 34 | 15 | 6 | 2 | 8 | 2 | 11 | 7
  Reticulocytes, changes to normal or no changes | 8 | 1 | 11 | 13 | 3 | 6 | 4 | 2 | 0 | 3 | 1 | 3 | 3
  Reticulocytes, increases to high: number analyzed (Participants) | 22 | 16 | 28 | 32 | 26 | 34 | 15 | 6 | 2 | 8 | 2 | 11 | 7
  Reticulocytes, increases to high | 10 | 10 | 12 | 15 | 14 | 21 | 11 | 2 | 2 | 4 | 1 | 3 | 2

27. Secondary Outcome: Part 2: Number of Participants With Worst Case Change From Baseline in Coagulation Parameters
Description: Blood samples were collected for evaluation of coagulation parameters. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with 'decreases to low', 'changes to normal' or 'no changes from Baseline', and 'increases to high' values have been presented. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Baseline (Day 1) and up to 42 months
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC)
Number analyzed (Participants) | 22 | 16 | 28 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
Participants
  Partial Thromboplastin Time, decreases to low: number analyzed (Participants) | 12 | 11 | 19 | 35 | 18 | 20 | 15 | 5 | 2 | 4 | 0 | 9 | 7
  Partial Thromboplastin Time, decreases to low | 2 | 0 | 3 | 0 | 0 | 1 | 2 | 0 | 1 | 0 |  | 0 | 1
  Partial Thromboplastin Time, changes to normal or no changes: number analyzed (Participants) | 12 | 11 | 19 | 35 | 18 | 20 | 15 | 5 | 2 | 4 | 0 | 9 | 7
  Partial Thromboplastin Time, changes to normal or no changes | 3 | 7 | 14 | 19 | 12 | 7 | 8 | 2 | 0 | 1 |  | 4 | 3
  Partial Thromboplastin Time, increases to high: number analyzed (Participants) | 12 | 11 | 19 | 35 | 18 | 20 | 15 | 5 | 2 | 4 | 0 | 9 | 7
  Partial Thromboplastin Time, increases to high | 8 | 4 | 2 | 16 | 6 | 12 | 6 | 3 | 1 | 3 |  | 5 | 3
  Prothrombin Intl. Normalized Ratio, decreases to low | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin Intl. Normalized Ratio, changes to normal or no changes | 17 | 2 | 23 | 24 | 18 | 15 | 8 | 5 | 2 | 8 | 2 | 9 | 6
  Prothrombin Intl. Normalized Ratio, increases to high | 5 | 14 | 5 | 13 | 10 | 18 | 8 | 1 | 0 | 0 | 0 | 2 | 1
  Prothrombin Time, decreases to low: number analyzed (Participants) | 22 | 15 | 26 | 37 | 27 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
  Prothrombin Time, decreases to low | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1
  Prothrombin Time, changes to normal or no changes: number analyzed (Participants) | 22 | 15 | 26 | 37 | 27 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
  Prothrombin Time, changes to normal or no changes | 9 | 5 | 18 | 16 | 14 | 17 | 7 | 2 | 1 | 4 | 2 | 6 | 4
  Prothrombin Time, increases to high: number analyzed (Participants) | 22 | 15 | 26 | 37 | 27 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
  Prothrombin Time, increases to high | 13 | 10 | 8 | 21 | 13 | 17 | 8 | 3 | 1 | 4 | 0 | 5 | 2

28. Secondary Outcome: Part 2: Number of Participants With Worst Case Change From Baseline in Urinalysis Parameters
Description: Urine samples were collected for evaluation of urinalysis parameters. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with 'decreases to low', 'changes to normal' or 'no changes from Baseline', and 'increases to high' values have been presented.
Time Frame: Baseline (Day 1) and up to 42 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC)
Number analyzed (Participants) | 22 | 16 | 28 | 37 | 28 | 34 | 16 | 5 | 2 | 8 | 2 | 9 | 7
Participants
  Occult Blood, No Change or Change to Negative | 19 | 10 | 20 | 28 | 18 | 20 | 13 | 3 | 2 | 5 | 2 | 3 | 4
  Occult Blood, Change to Positive | 3 | 6 | 8 | 9 | 10 | 14 | 3 | 2 | 0 | 3 | 0 | 6 | 3
  Protein, No Change or Change to Negative | 13 | 9 | 15 | 24 | 14 | 17 | 9 | 2 | 0 | 5 | 2 | 4 | 5
  Protein, Change to Positive | 9 | 7 | 13 | 13 | 14 | 17 | 7 | 3 | 2 | 3 | 0 | 5 | 2
  Ketones, No Change or Change to Negative | 17 | 9 | 22 | 27 | 20 | 24 | 9 | 4 | 2 | 8 | 2 | 7 | 4
  Ketones, Change to Positive | 5 | 7 | 6 | 10 | 8 | 10 | 7 | 1 | 0 | 0 | 0 | 2 | 3
  Glucose, No Change or Change to Negative | 20 | 15 | 24 | 32 | 24 | 34 | 14 | 5 | 2 | 7 | 2 | 9 | 7
  Glucose, Change to Positive | 2 | 1 | 4 | 5 | 4 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0

29. Secondary Outcome: Part 2: Changes From Baseline in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected from participants to assess urine pH levels.
Time Frame: Baseline (Day 1) and up to week 184
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Potential of Hydrogen (pH)
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC)
Number analyzed (Participants) | 22 | 16 | 29 | 36 | 28 | 34 | 15 | 5 | 2 | 8 | 2 | 9 | 7
Potential of Hydrogen (pH)
  Baseline: number analyzed (Participants) | 22 | 16 | 29 | 36 | 28 | 34 | 14 | 5 | 2 | 8 | 2 | 9 | 7
  Baseline | 5.95 (0.800) | 6.19 (0.772) | 5.97 (0.706) | 6.35 (0.715) | 6.00 (0.707) | 6.15 (0.784) | 6.36 (0.842) | 5.90 (0.224) | 5.75 (0.354) | 6.25 (0.845) | 5.50 (0.000) | 6.17 (0.707) | 5.43 (0.345)
  CFB to Day 8: number analyzed (Participants) | 21 | 15 | 26 | 36 | 28 | 34 | 13 | 4 | 1 | 7 | 2 | 9 | 7
  CFB to Day 8 | 0.07 (0.795) | -0.13 (0.694) | -0.15 (0.525) | -0.24 (0.760) | -0.04 (0.693) | -0.15 (0.892) | -0.19 (0.693) | -0.13 (0.250) | -0.50 (NA) — SD could not be calculated for single participant. | -0.21 (0.859) | 0.00 (0.000) | -0.06 (0.464) | 0.07 (0.189)
  CFB to Day 15: number analyzed (Participants) | 21 | 16 | 22 | 35 | 25 | 30 | 15 | 5 | 2 | 8 | 2 | 9 | 7
  CFB to Day 15 | 0.17 (0.842) | -0.16 (0.700) | 0.11 (0.706) | 0.01 (0.809) | -0.02 (0.620) | 0.03 (0.730) | 0.07 (0.842) | 0.10 (0.548) | 0.25 (0.354) | -0.25 (0.964) | 0.00 (0.707) | 0.06 (0.464) | 0.00 (0.577)
  CFB to Week 4 Day 1: number analyzed (Participants) | 17 | 16 | 18 | 35 | 24 | 30 | 13 | 5 | 2 | 5 | 2 | 9 | 7
  CFB to Week 4 Day 1 | -0.29 (0.902) | -0.06 (0.704) | -0.03 (0.899) | -0.23 (0.741) | -0.13 (0.837) | -0.32 (0.793) | -0.15 (0.966) | -0.20 (0.447) | 0.00 (0.707) | 0.00 (0.612) | 0.50 (0.707) | 0.33 (0.500) | -0.07 (0.189)
  CFB to Week 6 Day 1: number analyzed (Participants) | 14 | 13 | 16 | 30 | 24 | 30 | 15 | 4 | 1 | 5 | 1 | 7 | 6
  CFB to Week 6 Day 1 | 0.31 (0.727) | -0.54 (0.594) | -0.03 (0.591) | -0.42 (0.767) | 0.08 (0.929) | -0.48 (0.886) | -0.27 (0.942) | -0.13 (0.250) | 0.50 (NA) — SD could not be calculated for single participant. | -0.10 (0.822) | 0.50 (NA) — SD could not be calculated for single participant. | 0.14 (0.627) | 0.33 (0.606)
  CFB to Week 8: number analyzed (Participants) | 7 | 11 | 8 | 29 | 17 | 25 | 12 | 4 | 1 | 5 | 1 | 5 | 5
  CFB to Week 8 | 0.57 (1.018) | -0.50 (0.632) | -0.31 (0.651) | -0.16 (0.670) | -0.38 (0.944) | -0.30 (0.968) | -0.25 (0.783) | 0.13 (0.629) | 0.50 (NA) — SD could not be calculated for single participant. | 0.00 (0.935) | 0.00 (NA) — SD could not be calculated for single participant. | -0.10 (0.822) | 0.10 (0.224)
  CFB to Week 12: number analyzed (Participants) | 0 | 7 | 1 | 6 | 5 | 9 | 1 | 1 | 0 | 0 | 0 | 1 | 1
  CFB to Week 12 |  | 0.14 (0.988) | 0.00 (NA) — SD could not be calculated for single participant. | -0.17 (0.931) | 0.20 (0.837) | -0.33 (1.000) | -0.50 (NA) — SD could not be calculated for single participant. | -1.00 (NA) — SD could not be calculated for single participant. |  |  |  | 0.50 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 16: number analyzed (Participants) | 1 | 5 | 2 | 11 | 10 | 20 | 8 | 1 | 0 | 3 | 0 | 0 | 2
  CFB to Week 16 | -1.00 (NA) — SD could not be calculated for single participant. | -0.50 (0.791) | -0.25 (0.354) | 0.23 (0.932) | 0.10 (0.568) | -0.23 (1.032) | 0.31 (0.704) | -0.50 (NA) — SD could not be calculated for single participant. |  | -0.17 (0.764) |  |  | 0.75 (1.061)
  CFB to Week 20: number analyzed (Participants) | 0 | 4 | 0 | 4 | 1 | 8 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 20 |  | 0.00 (0.816) |  | 0.25 (0.866) | -0.50 (NA) — SD could not be calculated for single participant. | -0.19 (0.799) | 0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |
  CFB to Week 24: number analyzed (Participants) | 2 | 6 | 1 | 6 | 2 | 16 | 6 | 0 | 0 | 2 | 0 | 1 | 2
  CFB to Week 24 | -0.75 (0.354) | 0.00 (0.707) | 0.00 (NA) — SD could not be calculated for single participant. | 0.58 (1.201) | 0.25 (0.354) | -0.66 (1.012) | -0.67 (0.606) |  |  | 0.75 (1.061) |  | 0.50 (NA) — SD could not be calculated for single participant. | 0.00 (0.000)
  CFB to Week 28: number analyzed (Participants) | 0 | 4 | 0 | 2 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 28 |  | -0.13 (0.854) |  | 1.25 (0.354) |  | -0.75 (1.258) | 0.25 (0.354) |  |  |  |  |  |
  CFB to Week 32: number analyzed (Participants) | 1 | 3 | 0 | 3 | 2 | 13 | 4 | 1 | 0 | 1 | 0 | 0 | 2
  CFB to Week 32 | -0.50 (NA) — SD could not be calculated for single participant. | 0.00 (0.866) |  | 0.67 (0.577) | 0.25 (0.354) | -0.62 (1.121) | -0.25 (0.645) | 0.00 |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  | 0.00 (0.000)
  CFB to Week 36: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 36 | -0.50 (NA) — SD could not be calculated for single participant. | -0.17 (0.764) |  |  |  | -0.20 (0.570) |  |  |  |  |  |  |
  CFB to Week 40: number analyzed (Participants) | 1 | 2 | 0 | 2 | 0 | 13 | 4 | 0 | 0 | 0 | 0 | 0 | 2
  CFB to Week 40 | -1.00 (NA) — SD could not be calculated for single participant. | 0.25 (1.061) |  | 1.25 (1.061) |  | -0.54 (0.946) | -0.13 (0.629) |  |  |  |  |  | 0.00 (0.000)
  CFB to Week 44: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 44 | -1.50 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  | 0.50 (0.866) | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |
  CFB to Week 48: number analyzed (Participants) | 0 | 2 | 0 | 2 | 2 | 10 | 4 | 1 | 0 | 0 | 0 | 0 | 2
  CFB to Week 48 |  | 0.50 (1.414) |  | 1.00 (1.414) | 0.00 (0.000) | -0.50 (1.027) | -0.13 (0.629) | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.00 (0.000)
  CFB to Week 52: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 52 |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  | 0.38 (0.629) | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |
  CFB to Week 56: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 1
  CFB to Week 56 |  | 0.00 (NA) — SD could not be calculated for single participant. |  | 0.00 (NA) — SD could not be calculated for single participant. |  | -0.20 (0.570) | 0.00 (0.000) |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 60: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 60 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  | 0.50 (0.707) |  |  |  |  |  |  |
  CFB to Week 64: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 1
  CFB to Week 64 |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  | -0.50 (0.447) | -0.50 (0.707) |  |  |  |  |  | 0.00
  CFB to Week 68: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 68 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  | 0.25 (0.354) |  |  |  |  |  |  |
  CFB to Week 72: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 6 | 2 | 1 | 0 | 0 | 0 | 0 | 1
  CFB to Week 72 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  | -0.50 (0.707) | 0.00 (0.000) | 0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 76: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 76 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  | 0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |
  CFB to Week 80: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 80 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  | -0.38 (0.479) | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 84: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 84 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  | 2.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |
  CFB to Week 88: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 88 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  | -0.30 (0.671) | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |
  CFB to Week 92: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 92 |  | -1.00 (NA) — SD could not be calculated for single participant. |  |  |  | 1.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |
  CFB to Week 96: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 96 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  | 0.17 (1.443) |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 100: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 100 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 104: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 104 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  | -1.25 (0.354) |  |  |  |  |  |  |
  CFB to Week 108: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 108 |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 112: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 112 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 116: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 116 |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 120: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 120 |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 124: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 124 |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 128: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 128 |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 132: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 132 |  | 0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 136: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 136 |  |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 144: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 144 |  |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 152: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 152 |  |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 160: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 160 |  |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 168 |  |  |  |  |  |  |  | -0.50 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 176: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 176 |  |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 184: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 184 |  |  |  |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |

30. Secondary Outcome: Part 2: Changes From Baseline in Urine Specific Gravity
Description: Urine samples were collected from participants to assess urine specific gravity.
Time Frame: Baseline (Day 1) and up to week 184
Population: All treated population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC)
Number analyzed (Participants) | 22 | 16 | 29 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
Ratio
  Baseline: number analyzed (Participants) | 22 | 16 | 29 | 37 | 28 | 34 | 14 | 5 | 2 | 8 | 2 | 9 | 7
  Baseline | 1.02 (0.007) | 1.02 (0.006) | 1.02 (0.007) | 1.02 (0.007) | 1.02 (0.006) | 1.02 (1.02) | 1.02 (0.007) | 1.02 (0.012) | 1.02 (0.004) | 1.02 (0.007) | 1.03 (0.004) | 1.02 (0.007) | 1.02 (0.009)
  CFB to Day 8: number analyzed (Participants) | 21 | 15 | 26 | 37 | 28 | 33 | 13 | 4 | 1 | 7 | 2 | 9 | 7
  CFB to Day 8 | 0.00 (0.007) | 0.00 (0.008) | 0.00 (0.008) | 0.00 (0.007) | 0.00 (0.006) | 0.00 (0.007) | 0.00 (0.007) | 0.00 (0.003) | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.008) | 0.00 (0.000) | 0.00 (0.00) | 0.00 (0.005)
  CFB to Day 15: number analyzed (Participants) | 21 | 16 | 22 | 35 | 25 | 30 | 14 | 5 | 2 | 8 | 2 | 9 | 7
  CFB to Day 15 | 0.00 (0.007) | 0.00 (0.006) | 0.00 (0.005) | 0.00 (0.006) | 0.00 (0.006) | 0.00 (0.006) | 0.00 (0.008) | 0.00 (0.006) | 0.00 (0.004) | 0.00 (0.007) | 0.00 (0.000) | 0.00 (0.005) | 0.00 (0.006)
  CFB to Week 4 Day 1: number analyzed (Participants) | 17 | 16 | 18 | 34 | 24 | 30 | 13 | 5 | 2 | 5 | 2 | 9 | 7
  CFB to Week 4 Day 1 | 0.00 (0.007) | 0.00 (0.006) | 0.00 (0.006) | 0.00 (0.008) | 0.00 (0.007) | 0.00 (0.008) | 0.00 (0.009) | 0.00 (0.008) | 0.00 (0.000) | 0.00 (0.006) | -0.01 (0.004) | 0.00 (0.005) | 0.00 (0.006)
  CFB to Week 6 Day 1: number analyzed (Participants) | 14 | 13 | 16 | 30 | 24 | 30 | 15 | 4 | 1 | 5 | 1 | 7 | 6
  CFB to Week 6 Day 1 | 0.00 (0.008) | 0.00 (0.005) | 0.00 (0.006) | 0.00 (0.008) | 0.00 (0.008) | 0.00 (0.008) | 0.00 (0.010) | 0.01 (0.004) | -0.01 (NA) — SD could not be calculated for single participant. | 0.01 (0.005) | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.004) | 0.00 (0.010)
  CFB to Week 8: number analyzed (Participants) | 7 | 11 | 8 | 29 | 17 | 25 | 12 | 4 | 1 | 5 | 1 | 5 | 5
  CFB to Week 8 | 0.00 (0.008) | 0.00 (0.006) | 0.00 (0.008) | 0.00 (0.029) | 0.00 (0.007) | 0.00 (0.008) | 0.00 (0.009) | 0.00 (0.011) | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.003) | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.007) | 0.01 (0.005)
  CFB to Week 12: number analyzed (Participants) | 0 | 7 | 1 | 6 | 5 | 9 | 1 | 1 | 0 | 0 | 0 | 1 | 1
  CFB to Week 12 |  | 0.00 (0.005) | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.006) | 0.00 (0.011) | 0.00 (0.006) | -0.02 (NA) — SD could not be calculated for single participant. | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  | 0.00 (NA) — SD could not be calculated for single participant. | 0.01 (NA) — SD could not be calculated for single participant.
  CFB to Week 16: number analyzed (Participants) | 1 | 5 | 2 | 11 | 10 | 20 | 8 | 1 | 0 | 3 | 0 | 0 | 2
  CFB to Week 16 | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.008) | 0.00 (0.004) | 0.00 (0.007) | 0.00 (0.006) | 0.00 (0.009) | 0.01 (0.007) | 0.02 (NA) — SD could not be calculated for single participant. |  | 0.01 (0.005) |  |  | 0.01 (0.006)
  CFB to Week 20: number analyzed (Participants) | 0 | 4 | 0 | 4 | 1 | 8 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 20 |  | 0.00 (0.005) |  | 0.00 (0.010) | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.009) | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |
  CFB to Week 24: number analyzed (Participants) | 2 | 6 | 1 | 6 | 2 | 15 | 6 | 0 | 0 | 2 | 0 | 1 | 2
  CFB to Week 24 | 0.00 (0.002) | 0.00 (0.005) | 0.00 (NA) — SD could not be calculated for single participant. | NA (0.009) — SD could not be calculated for single participant. | 0.01 (0.011) | 0.00 (0.011) | 0.00 (0.007) |  |  | 0.00 (0.000) |  | -0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.001)
  CFB to Week 28: number analyzed (Participants) | 0 | 4 | 0 | 2 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 28 |  | 0.00 (0.008) |  | -0.01 (0.021) |  | 0.00 (0.015) | 0.00 (0.023) |  |  |  |  |  |
  CFB to Week 32: number analyzed (Participants) | 1 | 3 | 0 | 3 | 2 | 13 | 4 | 1 | 0 | 1 | 0 | 0 | 2
  CFB to Week 32 | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.005) |  | 0.00 (0.008) | 0.00 (0.000) | 0.00 (0.012) | 0.00 (0.011) | 0.02 (NA) — SD could not be calculated for single participant. |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  | 0.00 (0.007)
  CFB to Week 36: number analyzed (Participants) | 1 | 3 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 36 | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.003) |  |  |  | 0.01 (0.009) |  |  |  |  |  |  |
  CFB to Week 40: number analyzed (Participants) | 1 | 2 | 0 | 2 | 0 | 13 | 4 | 0 | 0 | 0 | 0 | 0 | 2
  CFB to Week 40 | 0.00 (NA) — SD could not be calculated for single participant. | -0.01 (0.007) |  | 0.00 (0.006) |  | 0.00 (0.011) | 0.01 (0.011) |  |  |  |  |  | -0.01 (0.011)
  CFB to Week 44: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 44 | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  | 0.00 (0.008) | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |
  CFB to Week 48: number analyzed (Participants) | 0 | 2 | 0 | 2 | 2 | 10 | 4 | 1 | 0 | 0 | 0 | 0 | 2
  CFB to Week 48 |  | -0.01 (0.000) |  | 0.01 (0.013) | 0.01 (0.011) | 0.01 (0.009) | 0.01 (0.013) | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.00 (0.002)
  CFB to Week 52: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 52 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  | 0.00 (0.008) | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |
  CFB to Week 56: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 1
  CFB to Week 56 |  | -0.01 (NA) — SD could not be calculated for single participant. |  | -0.01 (NA) — SD could not be calculated for single participant. |  | -0.01 (0.005) | 0.01 (0.009) |  |  |  |  |  | 0.01 (NA) — SD could not be calculated for single participant.
  CFB to Week 60: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 60 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  | -0.01 (0.001) |  |  |  |  |  |  |
  CFB to Week 64: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 1
  CFB to Week 64 |  |  |  | 0.01 (NA) — SD could not be calculated for single participant. |  | 0.00 (0.009) | 0.00 (0.011) |  |  |  |  |  | 0.01 (NA) — SD could not be calculated for single participant.
  CFB to Week 68: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 68 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  | -0.01 (0.002) |  |  |  |  |  |  |
  CFB to Week 72: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 5 | 2 | 1 | 0 | 0 | 0 | 0 | 1
  CFB to Week 72 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  | 0.00 (0.005) | 0.00 (0.001) | 0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  | 0.00 (NA) — SD could not be calculated for single participant.
  CFB to Week 76: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 76 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |
  CFB to Week 80: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 80 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  | 0.00 (0.004) | 0.00 (NA) — SD could not be calculated for single participant. | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 84: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 84 |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |
  CFB to Week 88: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 88 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  | 0.00 (0.005) | 0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |
  CFB to Week 92: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 92 |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |
  CFB to Week 96: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 96 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  | 0.00 (0.017) |  | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 100: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 100 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 104: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 104 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  | 0.00 (0.004) |  |  |  |  |  |  |
  CFB to Week 108: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 108 |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 112: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 112 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 116: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 116 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 120: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 120 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 124: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 124 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 128: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 128 |  | -0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 132: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CFB to Week 132 |  | 0.00 (NA) — SD could not be calculated for single participant. |  |  |  |  |  |  |  |  |  |  |
  CFB to Week 136: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 136 |  |  |  |  |  |  |  | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 144: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 144 |  |  |  |  |  |  |  | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 152: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 152 |  |  |  |  |  |  |  | 0.01 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 160: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 160 |  |  |  |  |  |  |  | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 168 |  |  |  |  |  |  |  | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 176: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 176 |  |  |  |  |  |  |  | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  |
  CFB to Week 184: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  CFB to Week 184 |  |  |  |  |  |  |  | 0.02 (NA) — SD could not be calculated for single participant. |  |  |  |  |

31. Secondary Outcome: Part 2: Number of Participants With Maximum Grade Worst Case Increase Post-baseline Relative to Baseline in Vital Signs
Description: The abnormal vital sign ranges are: Heart Rate:- Low (<60 beats per minute (bpm)), Normal (>=60 bpm to <=100 bpm), High (>100 bpm); Temperature:- Low (<=35 degree Celsius (C)), Normal (>35 C and <38 C), High (>=38 C); Systolic Blood Pressure:- Low (<90 millimeter of mercury (mmHg)), Normal (>=90 mmHg to <120 mmHg), High (>=120 mmHg); Diastolic Blood Pressure:- Low (<60 mmHg), Normal (>=60 mmHg to <80 mmHg), High (>=80 mmHg). Participants were counted in the worst-case category and their value changes to (low, normal or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Baseline (Day 1) and up to 42 months
Population: All treated population. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC)
Number analyzed (Participants) | 22 | 16 | 28 | 37 | 28 | 34 | 16 | 6 | 2 | 8 | 2 | 11 | 7
Participants
  Heart Rate, changes to low | 0 | 3 | 2 | 3 | 2 | 6 | 3 | 0 | 0 | 1 | 0 | 2 | 0
  Heart Rate, changes to normal or no changes | 14 | 5 | 25 | 19 | 17 | 21 | 7 | 4 | 1 | 6 | 2 | 7 | 5
  Heart Rate, changes to high | 8 | 9 | 1 | 16 | 9 | 8 | 6 | 2 | 1 | 1 | 0 | 3 | 2
  Temperature, changes to low | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Temperature, changes to normal or no changes | 21 | 14 | 28 | 36 | 25 | 31 | 16 | 4 | 2 | 8 | 2 | 10 | 7
  Temperature, changes to high | 1 | 2 | 0 | 0 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Systolic Blood Pressure, changes to low | 4 | 3 | 0 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1
  Systolic Blood Pressure, changes to normal or no changes | 14 | 7 | 20 | 28 | 21 | 23 | 12 | 5 | 1 | 7 | 2 | 8 | 4
  Systolic Blood Pressure, changes to high | 5 | 6 | 8 | 9 | 5 | 9 | 2 | 1 | 1 | 1 | 0 | 3 | 2
  Diastolic Blood Pressure, changes to low | 7 | 6 | 2 | 16 | 5 | 10 | 6 | 3 | 0 | 3 | 0 | 3 | 2
  Diastolic Blood Pressure, changes to normal or no changes | 10 | 6 | 20 | 15 | 18 | 16 | 7 | 2 | 1 | 3 | 1 | 6 | 4
  Diastolic Blood Pressure, changes to high | 8 | 4 | 6 | 11 | 6 | 11 | 4 | 3 | 1 | 2 | 1 | 3 | 1

32. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of GSK3326595
Description: Blood samples were collected for pharmacokinetic (PK) analysis of GSK3326595. PK parameter was determined using standard non-compartmental methods.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours (h) post-dose; pre-dose on day 8; pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 h post-dose on day 15
Population: Pharmacokinetic (PK) population included all participants from the All Treated Population for whom a PK sample was obtained and analyzed. Only those participants with data available at specified time points have been analyzed. Data was not available for samples that were out of stability or lost in transit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/ millilitre (ng/mL)
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 0
Nanogram/ millilitre (ng/mL)
  Day 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 0
  Day 1 | 14.1 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 70.7 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 288 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 508 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 653 (40.2) | 853 (29.4) | 1340 (48.4) | 1860 (41.4) | 55.8 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 210 (61.2) | 240 (93.9) | 925 (35.6) |
  Day 15: number analyzed (Participants) | 0 | 1 | 1 | 1 | 7 | 3 | 16 | 2 | 1 | 7 | 5 | 2 | 0
  Day 15 |  | 40.9 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 192 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 796 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 812 (35.1) | 678 (12.4) | 1600 (63.7) | 2810 (19.4) | 85.0 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 173 (37.6) | 368 (29.8) | 822 (26.3) |

33. Secondary Outcome: Part 3: Maximum Observed Plasma Concentration (Cmax) of GSK3326595
Description: as for outcome 32
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h post-dose
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 9
ng/mL | 291 (112)

34. Secondary Outcome: Part 1: Area Under the Plasma Concentration-time Curve (AUC) Extrapolated From Time Zero to Infinity (AUC[0-inf]) of GSK3326595
Description: as for outcome 32
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Nanogram/ millilitre (h*ng/mL)
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 0
Hour*Nanogram/ millilitre (h*ng/mL) |  | 349 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 926 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 1710 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 3240 (25.3) | 3800 (27.2) | 6760 (32.2) | 9610 (27.0) | 282 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 916 (42.9) | 1260 (47.9) | 4250 (65.1) |

35. Secondary Outcome: Part 3: Area Under the Plasma Concentration-time Curve (AUC) Extrapolated From Time Zero to Infinity (AUC[0-inf]) of GSK3326595
Description: as for outcome 32
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h post-dose
Population: as for outcome 33
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 8
h*ng/mL | 1770 (62.9)

36. Secondary Outcome: Part 1: AUC From Time Zero to the Last Quantifiable Concentration After Dosing (AUC[0-t]) of GSK3326595
Description: as for outcome 32
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 h post-dose; pre-dose on day 8; pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 h post-dose on day 15
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 0
h*ng/mL
  Day 1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 0
  Day 1 |  | 249 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 858 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 1610 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 3090 (26.7) | 3690 (28.1) | 6560 (32.5) | 9380 (26.6) | 249 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 816 (46.0) | 1100 (54.6) | 3950 (63.0) |
  Day 15: number analyzed (Participants) | 0 | 1 | 1 | 1 | 7 | 3 | 15 | 2 | 1 | 7 | 5 | 2 | 0
  Day 15 |  | 215 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 600 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 2040 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 4180 (32.9) | 4140 (29.0) | 7960 (41.7) | 12900 (32.8) | 370 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 965 (43.7) | 2360 (52.2) | 4040 (0.580) |

37. Secondary Outcome: Part 3: AUC From Time Zero to the Last Quantifiable Concentration After Dosing (AUC[0-t]) of GSK3326595
Description: as for outcome 32
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h post-dose
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified categories have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 9
h*ng/mL | 1480 (68.5)

38. Secondary Outcome: Part 1: AUC Over the Dosing Interval Tau (AUC[0-tau]) of GSK3326595
Description: as for outcome 32
Time Frame: as for outcome 36
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 0
h*ng/mL
  Day 1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 0
  Day 1 |  | 331 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 924 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 1710 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 3120 (25.9) | 3730 (25.5) | 6600 (32.7) | 9360 (26.7) | 250 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 819 (46.0) | 1100 (56.4) | 3970 (63.7) |
  Day 15: number analyzed (Participants) | 0 | 1 | 1 | 1 | 7 | 3 | 14 | 2 | 1 | 7 | 5 | 2 | 0
  Day 15 |  | 278 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 664 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 2050 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 4190 (33.1) | 4140 (28.8) | 8770 (24.1) | 12900 (32.6) | 374 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 1010 (41.7) | 2360 (52.3) | 4050 (1.20) |

39. Secondary Outcome: Part 3: AUC Over the Dosing Interval Tau (AUC[0-tau]) of GSK3326595
Description: as for outcome 32
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h post-dose
Population: Pharmacokinetic (PK) population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 8
h*ng/mL | 1640 (64.6)

40. Secondary Outcome: Part 1: Terminal Phase Half-life (t1/2) of GSK3326595
Description: as for outcome 32
Time Frame: as for outcome 36
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 0
Hour
  Day 1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 0
  Day 1 |  | 5.58 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 2.66 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 2.32 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 4.82 (30.4) | 3.71 (48.5) | 4.46 (20.9) | 5.03 (7.25) | 2.91 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 3.28 (26.2) | 3.32 (37.4) | 2.60 (10.4) |
  Day 15: number analyzed (Participants) | 0 | 1 | 1 | 1 | 7 | 2 | 15 | 2 | 1 | 5 | 3 | 2 | 0
  Day 15 |  | 4.57 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 3.32 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 5.30 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 6.30 (19.1) | 6.68 (10.9) | 4.68 (33.1) | 5.71 (3.33) | 2.93 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 4.21 (32.8) | 4.59 (20.3) | 3.76 (31.1) |

41. Secondary Outcome: Part 3: Terminal Phase Half-life (t1/2) of GSK3326595
Description: as for outcome 32
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h post-dose
Population: Pharmacokinetic (PK) population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 8
Hour | 5.44 (55.8)

42. Secondary Outcome: Part 1: Oral Clearance (CL/F) of GSK3326595
Description: as for outcome 32
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h post-dose
Population: as for outcome 32
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre/ hour (L/h)
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 7 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 0
Litre/ hour (L/h) |  | 71.7 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 54.0 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 58.5 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 61.8 (25.3) | 79.0 (27.2) | 59.2 (32.2) | 62.4 (27.0) | 355 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 218 (42.9) | 239 (47.9) | 94.1 (65.1) |

43. Secondary Outcome: Part 3: Oral Clearance (CL/F) of GSK3326595
Description: as for outcome 32
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h post-dose
Population: Pharmacokinetic (PK) population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 8
L/h | 56.4 (62.9)

44. Secondary Outcome: Part 1: Accumulation Ratio (AR) of GSK3326595
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h post-dose on Day 1 and Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h post-dose on Day 15
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified categories have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 7 | 3 | 14 | 2 | 1 | 7 | 5 | 2 | 0
Ratio |  | 0.840 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 0.719 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 1.20 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 1.34 (33.8) | 1.11 (8.37) | 1.34 (21.2) | 1.60 (23.3) | 1.50 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 1.23 (62.1) | 2.31 (38.1) | 1.43 (11.8) |

45. Secondary Outcome: Part 3: Accumulation Ratio (AR) of GSK3326595
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3326595
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h post-dose
Population: Pharmacokinetic (PK) population. Due to bioanalytical issues, PK data was not collected and analyzed. Therefore, this PK parameter was not reported in this study.
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 0

46. Secondary Outcome: Part 1: Time Invariance (TI) of GSK3326595
Description: Blood samples were collected for pharmacokinetic (PK) analysis of GSK3326595. PK parameter was determined using standard non-compartmental methods. Time invariance was calculated as AUC(0-tau) at Day 15 divided by AUC(0-infinity) at Day 1 for GSK3326595.
Time Frame: as for outcome 44
Population: Pharmacokinetic (PK) population.Only those participants with data available at specified categories have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 7 | 3 | 14 | 2 | 1 | 7 | 5 | 2 | 0
Ratio |  | 0.797 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 0.717 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 1.20 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 1.29 (32.7) | 1.09 (8.78) | 1.31 (20.8) | 1.56 (23.1) | 1.33 (NA) — Geometric Coefficient of Variation could not be calculated for single participant. | 1.10 (56.2) | 1.98 (33.7) | 1.34 (12.4) |

47. Secondary Outcome: Part 3: Time Invariance (TI) of GSK3326595
Description: Blood samples were collected for pharmacokinetic (PK) analysis of GSK3326595.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24h post-dose
Population: as for outcome 45
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 0

48. Secondary Outcome: Part 1: Overall Response Rate (ORR) Based on RECIST 1.1
Description: ORR was defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) per RECIST version 1.1. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm.
Time Frame: Up to 30 months
Population: All treated population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 8 | 3 | 19 | 3 | 1 | 7 | 6 | 3 | 15
Percentage of participants | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 25.0 [3.2 to 65.1] | 0 [0.0 to 70.8] | 5.3 [0.1 to 26.0] | 0 [0.0 to 70.8] | 0 [0.0 to 97.5] | 0 [0.0 to 41.0] | 0 [0.0 to 45.9] | 0 [0.0 to 70.8] | 6.7 [0.2 to 31.9]

49. Secondary Outcome: Part 2: Overall Response Rate (ORR) (Non-glioblastoma Multiforme [GBM] Cohorts)
Description: Overall response rate (ORR) was defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) per Response Evaluation Criteria in Solid Tumors Criteria (RECIST) version 1.1. Partial response (PR) was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response (CR) was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm).
Time Frame: Up to 42 months
Population: All treated population. Only participants in non-GBM cohorts were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 300mg (NSCLC)
Number analyzed (Participants) | 22 | 16 | 37 | 28 | 34 | 16 | 7
Percentage of participants | 0 [0.0 to 15.4] | 0 [0.0 to 20.6] | 2.7 [0.1 to 14.2] | 0 [0.0 to 12.3] | 2.9 [0.1 to 15.3] | 6.3 [0.2 to 30.2] | 0 [0.0 to 41.0]

50. Secondary Outcome: Part 2: Six-month Progression Free Survival (PFS) Rate (GBM Cohort)
Description: Six-month progression free survival (PFS) rate was defined as the percentage of participants free from radiographic progression per Response Assessment in Neuro-Oncology (RANO) criteria, or death due to any cause, for six months after starting GSK3326595. The RANO criteria were used to ascertain response (Wen, 2010).
Time Frame: At month 6
Population: All treated population. Only participants in GBM cohort was analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2: GSK3326595 400mg (GBM)
Number analyzed (Participants) | 29
Percentage of participants | 4 [0 to 17]

51. Secondary Outcome: Part 2: Duration of Response (DOR) (ACC Tablet Cohort)
Description: Duration of response (DOR) was defined as time from first evidence of response (CR or PR per RECIST 1.1) to earlier date of disease progression or death due to any cause, as determined by Investigator assessment.
Time Frame: Up to 42 months
Population: All treated population. Only participants with response in ACC tablets cohort were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: GSK3326595 300mg (ACC)
Number analyzed (Participants) | 1
Months | NA [NA to NA] — NA indicates that median and 95% confidence intervals could not be estimated due to insufficient number of participants with events and length of follow up in assessing the number of events.

52. Secondary Outcome: Part 3: ORR Based on Immune-based RECIST (iRECIST) Criteria
Description: ORR was defined as the percentage of participants with irCR or irPR per irRECIST. irCR is defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm). irPR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Up to 10 months
Population: All treated population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
Number analyzed (Participants) | 10
Percentage of participants | 0 [0.0 to 30.8]

53. Secondary Outcome: Part 2: ORR (GBM Cohort) Based on Response Assessment Neuro-Oncology (RANO) Working Group Criteria
Description: ORR was defined as the percentage of participants with a CR or PR, confirmed no less than 4 weeks based on the RANO criteria. CR was defined as complete disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks, stable or improved non-enhancing (T2/FLAIR) lesions, no new lesions, participants must be off corticosteroids (or on physiologic replacement doses only), and clinically stable or improved. PR was defined as at least 50% decrease compared to Baseline in the size of all measurable enhancing lesions sustained for at least 4 weeks, no progression of non-measurable disease or any new lesions, stable of lower dose of corticosteroids than Baseline dose, and stable or improved non-enhancing (T2/FLAIR) lesions.
Time Frame: Up to 42 months
Population: All treated population. Only participants in GBM cohort were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2: GSK3326595 400mg (GBM)
Number analyzed (Participants) | 29
Percentage of participants | 0 [0.0 to 11.9]

54. Secondary Outcome: Part 2: ORR (Non-Hodgkin's Lymphoma (NHL) Cohorts) Based on Lugano Criteria
Description: ORR was defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) based on Lugano Criteria for Non-Hodgkin's lymphoma cohorts.
Time Frame: Up to 42 months
Population: All treated population. Only participants in NHL cohorts were analyzed. For this analysis 300mg and 400 mg GSK3326595 arms were pooled based on NHL type to primarily serve the purpose for the comparison among the NHL cohorts.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Part 2: GSK3326595 400mg or 300mg (NHL P53 Mutant): Participant with non-Hodgkin's lymphoma (NHL) P53 Mutant received 400mg or 300 mg GSK3326595 capsules orally once a day.
- Part 2: GSK3326595 400mg or 300mg (NHL P53 Wild Type): Participant with NHL P53 Wild Type received 400 mg or 300mg GSK3326595 capsules orally once a day.
Arm/Group | Part 2: GSK3326595 400mg or 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg or 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown)
Number analyzed (Participants) | 8 | 10 | 11
Percentage of participants | 12.5 [0.3 to 52.7] | 10.0 [0.3 to 44.5] | 9.1 [0.2 to 41.3]

55. Secondary Outcome: Part 2: Overall Survival (OS) (ACC Tablet Cohort)
Description: Overall survival (OS) was defined as time from first dose until death from any cause in ACC participants who are systemic-treatment naïve.
Time Frame: Up to 42 months
Population: All treated population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: GSK3326595 300mg (ACC)
Number analyzed (Participants) | 16
Months | NA [NA to NA] — NA indicates that median and 95% confidence intervals could not be estimated due to insufficient number of participants with events and length of follow up in assessing the number of events.

56. Secondary Outcome: Part 2: Progression-free Survival
Description: PFS was defined as time from first dose until radiographic progression per standard criteria or death due to any cause, whichever is earlier.
Time Frame: Up to 42 months
Population: All treated population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 300mg (NSCLC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown)
Number analyzed (Participants) | 22 | 16 | 37 | 28 | 34 | 16 | 7 | 29 | 2 | 6 | 2 | 8 | 11
Months | 1.5 [1.5 to 1.8] | 3.6 [1.4 to 7.1] | 2.1 [1.6 to 4.2] | 3.2 [1.6 to 3.5] | 7.2 [4.8 to 11.0] | 7.1 [2.5 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants and length of follow-up in assessing the number of events. | 4.3 [1.4 to 17.9] | 1.3 [0.8 to 1.6] | 2.6 [NA to NA] — 95% CI was not estimable due to insufficient number of participants and length of follow-up in assessing the number of events. | 2.7 [1.7 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants and length of follow-up in assessing the number of events. | 2.6 [NA to NA] — 95% CI was not estimable due to insufficient number of participants and length of follow-up in assessing the number of events. | 4.5 [0.7 to 6.0] | 2.2 [1.1 to 3.7]

57. Secondary Outcome: RP2D Phase: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, or is a congenital anomaly/birth defect, other situations which involve medical or scientific judgment or was associated with liver injury and impaired liver function. SAEs are subset of AEs. AEs were coded using the MedDRA dictionary.
Time Frame: Up to maximum 42 months
Population: All treated population. For recommended phase 2 dose (RP2D) analysis, Part 1 and Part 2 arms were pooled based on dosage of GSK3326595.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 and Part 2: 400 QD Capsule (RP2D): Participant with relapsed and/or refractory solid tumors received 400 mg GSK3326595 capsules orally once a day at recommended phase 2 dose (RP2D) phase.
- Part 1 and Part 2: 300 QD Capsule (RP2D): Participant with relapsed and/or refractory solid tumors received 300 mg GSK3326595 capsules orally once a day at RP2D phase.
- Part 1 and Part 2: 300 QD Tablet (RP2D): Participant with relapsed and/or refractory solid tumors received 300 mg GSK3326595 tablets orally once a day at RP2D phase.
Arm/Group | Part 1 and Part 2: 400 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Tablet (RP2D)
Number analyzed (Participants) | 201 | 14 | 31
Participants
  Any AEs | 199 | 14 | 31
  Any SAEs | 92 | 3 | 11

58. Secondary Outcome: RP2D Phase: Number of Participants Withdrawn Due to AEs
Description: The data for number of participants withdrawn due to AEs have been presented.
Time Frame: Up to maximum 42 months
Population: as for outcome 57
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 and Part 2: 400 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Tablet (RP2D)
Number analyzed (Participants) | 201 | 14 | 31
Participants | 25 | 1 | 3

59. Secondary Outcome: RP2D Phase: Number of Participants With Dose Modifications of GSK3326595
Description: as for outcome 4
Time Frame: Up to maximum 42 months
Population: as for outcome 57
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 and Part 2: 400 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Tablet (RP2D)
Number analyzed (Participants) | 201 | 14 | 31
Participants
  Dose Interruptions | 127 | 9 | 27
  Dose Reductions | 123 | 6 | 11

60. Secondary Outcome: RP2D Phase: Number of Participants With Worst Case Change From Baseline in Clinical Chemistry Parameters
Description: as for outcome 25
Time Frame: Baseline (Day 1) and up to maximum 42 months
Population: All treated population. For recommended phase 2 dose (RP2D) analysis, Part 1 and Part 2 arms were pooled based on dosage of GSK3326595. Only those participants with data available at specified categories have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 and Part 2: 400 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Tablet (RP2D)
Number analyzed (Participants) | 200 | 14 | 31
Participants
  Alanine Aminotransferase, decreases to low | 15 | 1 | 11
  Alanine Aminotransferase, changes to normal or no changes | 165 | 11 | 20
  Alanine Aminotransferase, increases to high | 21 | 2 | 0
  Albumin, decreases to low | 80 | 1 | 14
  Albumin, changes to normal or no changes | 119 | 13 | 17
  Albumin, increases to high | 1 | 0 | 0
  Alkaline Phosphatase, decreases to low | 1 | 0 | 0
  Alkaline Phosphatase, changes to normal or no changes | 162 | 9 | 25
  Alkaline Phosphatase, increases to high | 37 | 5 | 6
  Amylase, decreases to low | 12 | 2 | 3
  Amylase, changes to normal or no changes | 166 | 12 | 27
  Amylase, increases to high | 23 | 0 | 1
  Aspartate Aminotransferase, decreases to low | 3 | 0 | 1
  Aspartate Aminotransferase, changes to normal or no changes | 147 | 10 | 26
  Aspartate Aminotransferase, increases to high | 50 | 4 | 4
  Bilirubin, decreases to low | 2 | 1 | 1
  Bilirubin, changes to normal or no changes | 164 | 12 | 24
  Bilirubin, increases to high | 34 | 1 | 6
  Calcium, decreases to low | 72 | 6 | 10
  Calcium, changes to normal or no changes | 122 | 8 | 21
  Calcium, increases to high | 8 | 0 | 0
  Creatinine, decreases to low | 26 | 2 | 6
  Creatinine, changes to normal or no changes | 138 | 11 | 23
  Creatinine, increases to high | 36 | 1 | 3
  Direct Bilirubin, decreases to low: number analyzed (Participants) | 199 | 14 | 31
  Direct Bilirubin, decreases to low | 0 | 0 | 0
  Direct Bilirubin, changes to normal or no changes: number analyzed (Participants) | 199 | 14 | 31
  Direct Bilirubin, changes to normal or no changes | 129 | 10 | 19
  Direct Bilirubin, increases to high: number analyzed (Participants) | 199 | 14 | 31
  Direct Bilirubin, increases to high | 70 | 4 | 12
  Glucose, decreases to low | 14 | 2 | 3
  Glucose, changes to normal or no changes | 120 | 9 | 20
  Glucose, increases to high | 70 | 3 | 9
  Lipase, decreases to low | 8 | 1 | 3
  Lipase, changes to normal or no changes | 165 | 10 | 28
  Lipase, increases to high | 28 | 3 | 0
  Potassium, decreases to low | 24 | 2 | 6
  Potassium, changes to normal or no changes | 142 | 8 | 21
  Potassium, increases to high | 39 | 4 | 4
  Protein, decreases to low | 77 | 5 | 13
  Protein, changes to normal or no changes | 116 | 9 | 17
  Protein, increases to high | 8 | 0 | 1
  Sodium, decreases to low | 39 | 2 | 6
  Sodium, changes to normal or no changes | 149 | 12 | 21
  Sodium, increases to high | 14 | 0 | 4
  Urea Nitrogen, decreases to low: number analyzed (Participants) | 92 | 4 | 29
  Urea Nitrogen, decreases to low | 5 | 0 | 3
  Urea Nitrogen, changes to normal or no changes: number analyzed (Participants) | 92 | 4 | 29
  Urea Nitrogen, changes to normal or no changes | 53 | 3 | 17
  Urea Nitrogen, increases to high: number analyzed (Participants) | 92 | 4 | 29
  Urea Nitrogen, increases to high | 36 | 1 | 9

61. Secondary Outcome: RP2D Phase: Number of Participants With Worst Case Change From Baseline in Hematology Parameters
Description: Blood samples were collected for evaluation of hematology parameters. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v5.0. The number of participants with 'decreases to low', 'changes to normal' or 'no changes from Baseline', and 'increases to high' values have been presented. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Baseline (Day 1) and up to maximum 42 months
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 and Part 2: 400 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Tablet (RP2D)
Number analyzed (Participants) | 200 | 14 | 31
Participants
  Basophils, decreases to low: number analyzed (Participants) | 190 | 14 | 31
  Basophils, decreases to low | 5 | 0 | 0
  Basophils, changes to normal or no changes: number analyzed (Participants) | 190 | 14 | 31
  Basophils, changes to normal or no changes | 183 | 13 | 31
  Basophils, increases to high: number analyzed (Participants) | 190 | 14 | 31
  Basophils, increases to high | 3 | 1 | 0
  Eosinophils, decreases to low: number analyzed (Participants) | 190 | 14 | 31
  Eosinophils, decreases to low | 12 | 0 | 3
  Eosinophils, changes to normal or no changes: number analyzed (Participants) | 190 | 14 | 31
  Eosinophils, changes to normal or no changes | 170 | 11 | 28
  Eosinophils, increases to high: number analyzed (Participants) | 190 | 14 | 31
  Eosinophils, increases to high | 8 | 3 | 1
  Mean Corpuscular Hemoglobin, decreases to low: number analyzed (Participants) | 199 | 14 | 31
  Mean Corpuscular Hemoglobin, decreases to low | 18 | 0 | 8
  Mean Corpuscular Hemoglobin, changes to normal or no changes: number analyzed (Participants) | 199 | 14 | 31
  Mean Corpuscular Hemoglobin, changes to normal or no changes | 173 | 14 | 21
  Mean Corpuscular Hemoglobin, increases to high: number analyzed (Participants) | 199 | 14 | 31
  Mean Corpuscular Hemoglobin, increases to high | 8 | 0 | 2
  Mean Corpuscular Volume, decreases to low | 14 | 0 | 0
  Mean Corpuscular Volume, changes to normal or no changes | 173 | 13 | 28
  Mean Corpuscular Volume, increases to high | 13 | 1 | 3
  Erythrocytes, decreases to low: number analyzed (Participants) | 199 | 14 | 31
  Erythrocytes, decreases to low | 94 | 7 | 17
  Erythrocytes, changes to normal or no changes: number analyzed (Participants) | 199 | 14 | 31
  Erythrocytes, changes to normal or no changes | 104 | 7 | 13
  Erythrocytes, increases to high: number analyzed (Participants) | 199 | 14 | 31
  Erythrocytes, increases to high | 1 | 1 | 1
  Hematocrit, decreases to low | 108 | 9 | 15
  Hematocrit, changes to normal or no changes | 92 | 5 | 16
  Hematocrit, increases to high | 0 | 0 | 0
  Hemoglobin, decreases to low | 106 | 10 | 16
  Hemoglobin, changes to normal or no changes | 94 | 4 | 15
  Hemoglobin, increases to high | 0 | 0 | 0
  Leukocytes, decreases to low | 93 | 5 | 16
  Leukocytes, changes to normal or no changes | 91 | 6 | 13
  Leukocytes, increases to high | 22 | 3 | 4
  Lymphocytes, decreases to low | 64 | 6 | 11
  Lymphocytes, changes to normal or no changes | 136 | 7 | 20
  Lymphocytes, increases to high | 0 | 1 | 0
  Monocytes, decreases to low: number analyzed (Participants) | 190 | 14 | 31
  Monocytes, decreases to low | 31 | 3 | 1
  Monocytes, changes to normal or no changes: number analyzed (Participants) | 190 | 14 | 31
  Monocytes, changes to normal or no changes | 129 | 8 | 21
  Monocytes, increases to high: number analyzed (Participants) | 190 | 14 | 31
  Monocytes, increases to high | 38 | 3 | 9
  Neutrophils, decreases to low | 59 | 6 | 9
  Neutrophils, changes to normal or no changes | 115 | 6 | 17
  Neutrophils, increases to high | 30 | 2 | 6
  Platelets, decreases to low | 110 | 5 | 12
  Platelets, changes to normal or no changes | 79 | 8 | 17
  Platelets, increases to high | 22 | 1 | 4
  Reticulocytes, decreases to low: number analyzed (Participants) | 193 | 14 | 30
  Reticulocytes, decreases to low | 86 | 3 | 9
  Reticulocytes, changes to normal or no changes: number analyzed (Participants) | 193 | 14 | 30
  Reticulocytes, changes to normal or no changes | 51 | 5 | 8
  Reticulocytes, increases to high: number analyzed (Participants) | 193 | 14 | 30
  Reticulocytes, increases to high | 97 | 7 | 19

62. Secondary Outcome: RP2D Phase: Number of Participants With Worst Case Change From Baseline in Coagulation Parameters
Description: as for outcome 27
Time Frame: Baseline (Day 1) and up to maximum 42 months
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 and Part 2: 400 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Tablet (RP2D)
Number analyzed (Participants) | 200 | 14 | 31
Participants
  Partial Thromboplastin Time, decreases to low: number analyzed (Participants) | 140 | 11 | 30
  Partial Thromboplastin Time, decreases to low | 6 | 2 | 3
  Partial Thromboplastin Time, changes to normal or no changes: number analyzed (Participants) | 140 | 11 | 30
  Partial Thromboplastin Time, changes to normal or no changes | 72 | 4 | 15
  Partial Thromboplastin Time, increases to high: number analyzed (Participants) | 140 | 11 | 30
  Partial Thromboplastin Time, increases to high | 63 | 5 | 13
  Prothrombin Intl. Normalized Ratio, decreases to low | 1 | 0 | 0
  Prothrombin Intl. Normalized Ratio, changes to normal or no changes | 125 | 12 | 13
  Prothrombin Intl. Normalized Ratio, increases to high | 74 | 2 | 18
  Prothrombin Time, decreases to low: number analyzed (Participants) | 194 | 14 | 31
  Prothrombin Time, decreases to low | 2 | 1 | 2
  Prothrombin Time, changes to normal or no changes: number analyzed (Participants) | 194 | 14 | 31
  Prothrombin Time, changes to normal or no changes | 95 | 10 | 14
  Prothrombin Time, increases to high: number analyzed (Participants) | 194 | 14 | 31
  Prothrombin Time, increases to high | 98 | 3 | 16

63. Secondary Outcome: RP2D Phase: Number of Participants With Worst Case Change From Baseline in Urinalysis Parameters
Description: Urine samples were collected for evaluation of urinalysis parameters. The summaries of worst case change from Baseline with respect to normal range have been presented for only those laboratory tests that are gradable by CTCAE v4.0. The number of participants with 'decreases to low', 'changes to normal' or 'no changes from Baseline', and 'increases to high' values have been presented.
Time Frame: Baseline (Day 1) and up to maximum 42 months
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 and Part 2: 400 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Tablet (RP2D)
Number analyzed (Participants) | 197 | 14 | 31
Participants
  Occult Blood, No Change or Change to Negative | 133 | 10 | 23
  Occult Blood, Change to Positive | 64 | 4 | 8
  Protein, No Change or Change to Negative | 110 | 9 | 19
  Protein, Change to Positive | 87 | 5 | 12
  Ketones, No Change or Change to Negative | 144 | 10 | 17
  Ketones, Change to Positive | 53 | 4 | 14
  Glucose, No Change or Change to Negative | 179 | 14 | 25
  Glucose, Change to Positive | 18 | 0 | 6

64. Secondary Outcome: RP2D Phase: Changes From Baseline in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected from participants to assess urine pH levels.
Time Frame: Baseline (Day 1) and up to Week 184
Population: All treated population. For recommended phase 2 dose (RP2D) analysis, Part 1 and Part 2 arms were pooled based on dosage of GSK3326595. Only those participants with data available at specified time point have been analyzed.
Measure: Mean (Standard Deviation); unit: Potential of Hydrogen (pH)
Arm/Group | Part 1 and Part 2: 400 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Tablet (RP2D)
Number analyzed (Participants) | 196 | 14 | 30
Potential of Hydrogen (pH)
  Baseline: number analyzed (Participants) | 196 | 14 | 29
  Baseline | 6.11 (0.729) | 5.64 (0.413) | 5.98 (0.901)
  CFB to Day 8: number analyzed (Participants) | 190 | 12 | 28
  CFB to Day 8 | -0.13 (0.711) | -0.04 (0.257) | -0.11 (0.599)
  CFB to Day 15: number analyzed (Participants) | 180 | 14 | 30
  CFB to Day 15 | 0.01 (0.722) | 0.00 (0.480) | 0.05 (0.770)
  CFB to Week 4 Day 1: number analyzed (Participants) | 166 | 13 | 28
  CFB to Week 4 Day 1 | -0.16 (0.769) | -0.08 (0.494) | -0.13 (0.888)
  CFB to Week 6 Day 1: number analyzed (Participants) | 149 | 10 | 27
  CFB to Week 6 Day 1 | -0.20 (0.807) | 0.30 (0.483) | -0.17 (0.899)
  CFB to Week 8: number analyzed (Participants) | 116 | 9 | 21
  CFB to Week 8 | -0.20 (0.823) | -0.06 (0.464) | 0.05 (0.805)
  CFB to Week 12: number analyzed (Participants) | 33 | 2 | 7
  CFB to Week 12 | -0.06 (0.873) | -0.25 (0.354) | 0.00 (0.957)
  CFB to Week 16: number analyzed (Participants) | 55 | 3 | 12
  CFB to Week 16 | -0.11 (0.859) | 0.50 (0.866) | 0.17 (0.615)
  CFB to Week 20: number analyzed (Participants) | 18 | 0 | 5
  CFB to Week 20 | -0.03 (0.757) |  | 0.00 (0.791)
  CFB to Week 24: number analyzed (Participants) | 37 | 2 | 11
  CFB to Week 24 | -0.15 (1.020) | 0.00 (0.000) | -0.64 (0.505)
  CFB to Week 28: number analyzed (Participants) | 11 | 0 | 7
  CFB to Week 28 | -0.05 (1.128) |  | -0.21 (0.488)
  CFB to Week 32: number analyzed (Participants) | 25 | 2 | 9
  CFB to Week 32 | -0.22 (0.980) | 0.00 (0.000) | -0.06 (0.950)
  CFB to Week 36: number analyzed (Participants) | 9 | 0 | 4
  CFB to Week 36 | -0.22 (0.565) |  | -0.63 (0.479)
  CFB to Week 40: number analyzed (Participants) | 18 | 2 | 9
  CFB to Week 40 | -0.28 (1.074) | 0.00 (0.000) | -0.17 (0.661)
  CFB to Week 44: number analyzed (Participants) | 5 | 0 | 5
  CFB to Week 44 | 0.00 (1.061) |  | -0.10 (0.742)
  CFB to Week 48: number analyzed (Participants) | 17 | 2 | 9
  CFB to Week 48 | -0.12 (1.068) | 0.00 (0.000) | -0.33 (0.661)
  CFB to Week 52: number analyzed (Participants) | 5 | 0 | 6
  CFB to Week 52 | 0.30 (0.570) |  | -0.25 (0.274)
  CFB to Week 56: number analyzed (Participants) | 7 | 1 | 6
  CFB to Week 56 | -0.14 (0.476) | 0.00 | -0.42 (0.492)
  CFB to Week 60: number analyzed (Participants) | 3 | 0 | 3
  CFB to Week 60 | 0.17 (0.764) |  | -1.00 (0.500)
  CFB to Week 64: number analyzed (Participants) | 7 | 1 | 5
  CFB to Week 64 | -0.43 (0.450) | 0.00 | -0.40 (0.652)
  CFB to Week 68: number analyzed (Participants) | 3 | 0 | 4
  CFB to Week 68 | 0.00 (0.500) |  | -0.25 (0.866)
  CFB to Week 72: number analyzed (Participants) | 8 | 1 | 5
  CFB to Week 72 | -0.38 (0.694) | 0.00 (NA) — SD could not be calculated for single participant. | -0.20 (0.570)
  CFB to Week 76: number analyzed (Participants) | 2 | 0 | 2
  CFB to Week 76 | 0.00 (0.707) |  | -0.75 (0.354)
  CFB to Week 80: number analyzed (Participants) | 6 | 0 | 4
  CFB to Week 80 | -0.33 (0.408) |  | 0.00 (0.707)
  CFB to Week 84: number analyzed (Participants) | 2 | 0 | 1
  CFB to Week 84 | 0.75 (1.768) |  | 0.00
  CFB to Week 88: number analyzed (Participants) | 6 | 0 | 3
  CFB to Week 88 | -0.33 (0.606) |  | -0.17 (0.764)
  CFB to Week 92: number analyzed (Participants) | 2 | 0 | 2
  CFB to Week 92 | 0.00 (1.414) |  | -0.75 (0.354)
  CFB to Week 96: number analyzed (Participants) | 5 | 0 | 3
  CFB to Week 96 | 0.00 (1.061) |  | -0.33 (0.289)
  CFB to Week 100: number analyzed (Participants) | 1 | 0 | 2
  CFB to Week 100 | -0.50 (NA) — SD could not be calculated for single participant. |  | -0.25 (0.354)
  CFB to Week 104: number analyzed (Participants) | 3 | 0 | 3
  CFB to Week 104 | -1.00 (0.500) |  | -0.83 (0.289)
  CFB to Week 108: number analyzed (Participants) | 1 | 0 | 2
  CFB to Week 108 | 0.00 (NA) — SD could not be calculated for single participant. |  | -1.00 (0.000)
  CFB to Week 112: number analyzed (Participants) | 2 | 0 | 3
  CFB to Week 112 | -0.50 (0.000) |  | -0.50 (0.866)
  CFB to Week 116: number analyzed (Participants) | 1 | 0 | 2
  CFB to Week 116 | 0.00 (NA) — SD could not be calculated for single participant. |  | -0.75 (0.354)
  CFB to Week 120: number analyzed (Participants) | 1 | 0 | 3
  CFB to Week 120 | 0.00 (NA) — SD could not be calculated for single participant. |  | -0.33 (0.289)
  CFB to Week 124: number analyzed (Participants) | 1 | 0 | 1
  CFB to Week 124 | 0.00 (NA) — SD could not be calculated for single participant. |  | -0.50 (NA) — SD could not be calculated for single participant.
  CFB to Week 128: number analyzed (Participants) | 1 | 0 | 3
  CFB to Week 128 | -0.50 (NA) — SD could not be calculated for single participant. |  | -0.33 (0.764)
  CFB to Week 132: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 132 | 0.50 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 136: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 136 | -0.50 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 144: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 144 | 0.00 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 152: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 152 | 0.00 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 160: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 160 | -0.50 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 168: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 168 | -0.50 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 176: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 176 | 0.00 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 184: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 184 | 0.00 (NA) — SD could not be calculated for single participant. |  |

65. Secondary Outcome: RP2D Phase: Changes From Baseline in Urine Specific Gravity
Description: Urine samples were collected from participants to assess urine specific gravity.
Time Frame: Baseline (Day 1) and up to Week 184
Population: All treated population. For recommended phase 2 dose (RP2D) analysis, Part 1 and Part 2 arms were pooled based on dosage of GSK3326595. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1 and Part 2: 400 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Tablet (RP2D)
Number analyzed (Participants) | 197 | 14 | 29
Ratio
  Baseline | 1.02 (0.007) | 1.02 (0.007) | 1.02 (0.007)
  CFB to Day 8: number analyzed (Participants) | 189 | 12 | 28
  CFB to Day 8 | 0.00 (0.007) | 0.00 (0.005) | 0.00 (0.008)
  CFB to Day 15: number analyzed (Participants) | 180 | 14 | 29
  CFB to Day 15 | 0.00 (0.006) | 0.00 (0.006) | 0.00 (0.008)
  CFB to Week 4 Day 1: number analyzed (Participants) | 165 | 13 | 28
  CFB to Week 4 Day 1 | 0.00 (0.007) | 0.00 (0.006) | 0.00 (0.008)
  CFB to Week 6 Day 1: number analyzed (Participants) | 149 | 10 | 27
  CFB to Week 6 Day 1 | 0.00 (0.007) | 0.00 (0.009) | 0.00 (0.008)
  CFB to Week 8: number analyzed (Participants) | 116 | 9 | 21
  CFB to Week 8 | 0.00 (0.016) | 0.00 (0.009) | 0.00 (0.008)
  CFB to Week 12: number analyzed (Participants) | 33 | 2 | 7
  CFB to Week 12 | 0.00 (0.007) | 0.00 (0.008) | 0.00 (0.008)
  CFB to Week 16: number analyzed (Participants) | 55 | 3 | 12
  CFB to Week 16 | 0.00 (0.008) | 0.00 (0.015) | 0.00 (0.007)
  CFB to Week 20: number analyzed (Participants) | 18 | 0 | 5
  CFB to Week 20 | 0.00 (0.008) |  | 0.00 (0.006)
  CFB to Week 24: number analyzed (Participants) | 36 | 2 | 11
  CFB to Week 24 | 0.00 (0.009) | 0.00 (0.001) | 0.00 (0.005)
  CFB to Week 28: number analyzed (Participants) | 11 | 0 | 7
  CFB to Week 28 | 0.00 (0.012) |  | 0.00 (0.010)
  CFB to Week 32: number analyzed (Participants) | 25 | 2 | 9
  CFB to Week 32 | 0.00 (0.010) | 0.00 (0.007) | 0.00 (0.007)
  CFB to Week 36: number analyzed (Participants) | 9 | 0 | 4
  CFB to Week 36 | 0.00 (0.008) |  | 0.00 (0.002)
  CFB to Week 40: number analyzed (Participants) | 18 | 2 | 9
  CFB to Week 40 | 0.00 (0.010) | -0.01 (0.011) | 0.00 (0.008)
  CFB to Week 44: number analyzed (Participants) | 5 | 0 | 5
  CFB to Week 44 | 0.00 (0.007) |  | 0.00 (0.007)
  CFB to Week 48: number analyzed (Participants) | 17 | 2 | 9
  CFB to Week 48 | 0.01 (0.010) | 0.00 (0.002) | 0.00 (0.009)
  CFB to Week 52: number analyzed (Participants) | 5 | 0 | 6
  CFB to Week 52 | 0.00 (0.008) |  | 0.00 (0.007)
  CFB to Week 56: number analyzed (Participants) | 6 | 1 | 6
  CFB to Week 56 | -0.01 (0.004) | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.008)
  CFB to Week 60: number analyzed (Participants) | 3 | 0 | 3
  CFB to Week 60 | -0.01 (0.004) |  | 0.00 (0.006)
  CFB to Week 64: number analyzed (Participants) | 6 | 1 | 5
  CFB to Week 64 | 0.00 (0.009) | 0.01 (NA) — SD could not be calculated for single participant. | 0.00 (0.008)
  CFB to Week 68: number analyzed (Participants) | 3 | 0 | 4
  CFB to Week 68 | -0.01 (0.002) |  | 0.00 (0.003)
  CFB to Week 72: number analyzed (Participants) | 7 | 1 | 5
  CFB to Week 72 | 0.00 (0.006) | 0.00 (NA) — SD could not be calculated for single participant. | 0.00 (0.001)
  CFB to Week 76: number analyzed (Participants) | 2 | 0 | 2
  CFB to Week 76 | -0.01 (0.004) |  | 0.00 (0.004)
  CFB to Week 80: number analyzed (Participants) | 6 | 0 | 4
  CFB to Week 80 | 0.00 (0.008) |  | 0.00 (0.005)
  CFB to Week 84: number analyzed (Participants) | 2 | 0 | 1
  CFB to Week 84 | -0.01 (0.008) |  | 0.00
  CFB to Week 88: number analyzed (Participants) | 6 | 0 | 3
  CFB to Week 88 | 0.00 (0.004) |  | 0.00 (0.005)
  CFB to Week 92: number analyzed (Participants) | 2 | 0 | 2
  CFB to Week 92 | 0.00 (0.006) |  | 0.00 (0.006)
  CFB to Week 96: number analyzed (Participants) | 5 | 0 | 3
  CFB to Week 96 | 0.00 (0.017) |  | 0.00 (0.003)
  CFB to Week 100: number analyzed (Participants) | 1 | 0 | 2
  CFB to Week 100 | -0.01 (NA) — SD could not be calculated for single participant. |  | 0.00 (0.001)
  CFB to Week 104: number analyzed (Participants) | 3 | 0 | 3
  CFB to Week 104 | 0.00 (0.003) |  | -0.01 (0.008)
  CFB to Week 108: number analyzed (Participants) | 1 | 0 | 2
  CFB to Week 108 | 0.00 (NA) — SD could not be calculated for single participant. |  | 0.00 (0.004)
  CFB to Week 112: number analyzed (Participants) | 2 | 0 | 3
  CFB to Week 112 | 0.01 (0.020) |  | 0.00 (0.007)
  CFB to Week 116: number analyzed (Participants) | 1 | 0 | 2
  CFB to Week 116 | -0.01 (NA) — SD could not be calculated for single participant. |  | 0.00 (0.004)
  CFB to Week 120: number analyzed (Participants) | 1 | 0 | 3
  CFB to Week 120 | -0.01 (NA) — SD could not be calculated for single participant. |  | 0.01 (0.008)
  CFB to Week 124: number analyzed (Participants) | 1 | 0 | 1
  CFB to Week 124 | -0.01 (NA) — SD could not be calculated for single participant. |  | 0.01 (NA) — SD could not be calculated for single participant.
  CFB to Week 128: number analyzed (Participants) | 1 | 0 | 3
  CFB to Week 128 | -0.01 (NA) — SD could not be calculated for single participant. |  | 0.01 (0.008)
  CFB to Week 132: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 132 | 0.00 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 136: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 136 | 0.02 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 144: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 144 | 0.02 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 152: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 152 | 0.01 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 160: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 160 | 0.02 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 168: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 168 | 0.02 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 176: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 176 | 0.02 (NA) — SD could not be calculated for single participant. |  |
  CFB to Week 184: number analyzed (Participants) | 1 | 0 | 0
  CFB to Week 184 | 0.02 (NA) — SD could not be calculated for single participant. |  |

66. Secondary Outcome: RP2D Phase: Number of Participants With Worst-case Increase Post-baseline Relative to Baseline in Vital Signs
Description: Vital signs were measured. The abnormal vital sign ranges are: Heart Rate:- Low [<60 beats per minute (bpm)], Normal (>=60 bpm to <=100 bpm), High (>100 bpm); Temperature:- Low (<=35 C), Normal (>35 C and <38 C), High (>=38 C); Systolic Blood Pressure:- Low (<90 mmHg), Normal (>=90 mmHg to <120 mmHg), High (>=120 mmHg); Diastolic Blood Pressure:- Low (<60 mmHg), Normal (>=60 mmHg to <80 mmHg), High (>=80 mmHg). Participants were counted in the worst-case category that their value changes to (low, normal or high), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Baseline (Day 1) and up to maximum 42 months
Population: as for outcome 60
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 and Part 2: 400 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Capsule (RP2D) | Part 1 and Part 2: 300 QD Tablet (RP2D)
Number analyzed (Participants) | 200 | 14 | 31
Participants
  Heart Rate, changes to low | 19 | 0 | 5
  Heart Rate, changes to normal or no changes | 124 | 11 | 17
  Heart Rate, changes to high | 61 | 3 | 9
  Temperature, changes to low | 2 | 0 | 0
  Temperature, changes to normal or no changes | 186 | 14 | 31
  Temperature, changes to high | 12 | 0 | 0
  Systolic Blood Pressure, changes to low | 14 | 1 | 4
  Systolic Blood Pressure, changes to normal or no changes | 139 | 9 | 23
  Systolic Blood Pressure, changes to high | 49 | 4 | 4
  Diastolic Blood Pressure, changes to low | 57 | 4 | 9
  Diastolic Blood Pressure, changes to normal or no changes | 101 | 7 | 15
  Diastolic Blood Pressure, changes to high | 57 | 4 | 9

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected up to 30 months for part 1, 42 months for part 2 and 10 months for part 3.
Description: All Treated population included all participants who received at least one dose of GSK3326595.
Arm/Group | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) | Part 1: GSK3326595 25mg QD | Part 1: GSK3326595 50mg QD | Part 1: GSK3326595 100mg QD | Part 1: GSK3326595 200mg QD | Part 1: GSK3326595 300mg QD | Part 1: GSK3326595 400mg QD | Part 1: GSK3326595 600mg QD | Part 1: GSK3326595 50mg Twice Daily (BID) | Part 1: GSK3326595 100mg BID | Part 1: GSK3326595 150mg BID | Part 1: GSK3326595 200mg BID | Part 1: GSK3326595 300mg QD (Food Effect) | Part 2: GSK3326595 400mg (TNBC) | Part 2: GSK3326595 400mg (mTCC) | Part 2: GSK3326595 400mg (GBM) | Part 2: GSK3326595 400mg (ER+BC) | Part 2: GSK3326595 400mg (HPV+) | Part 2: GSK3326595 400mg (ACC) | Part 2: GSK3326595 300mg (ACC) | Part 2: GSK3326595 400mg (NHL P53 Mutant) | Part 2: GSK3326595 300mg (NHL P53 Mutant) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) | Part 2: GSK3326595 400mg (NHL P53 Unknown) | Part 2: GSK3326595 300mg (NSCLC) | Part 3: GSK3326595 100mg + Pembrolizumab 200mg
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 0/1 | 7/8 | 3/3 | 13/19 | 3/3 | 1/1 | 6/7 | 6/6 | 3/3 | 8/15 | 16/22 | 10/16 | 22/29 | 31/37 | 25/28 | 20/34 | 2/16 | 4/6 | 1/2 | 5/8 | 1/2 | 7/11 | 3/7 | 6/10
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 4/8 | 1/3 | 10/19 | 1/3 | 0/1 | 2/7 | 3/6 | 3/3 | 6/15 | 13/22 | 7/16 | 15/29 | 10/37 | 13/28 | 15/34 | 5/16 | 4/6 | 2/2 | 4/8 | 0/2 | 4/11 | 0/7 | 5/10
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 7/8 | 3/3 | 19/19 | 3/3 | 1/1 | 7/7 | 6/6 | 3/3 | 15/15 | 22/22 | 16/16 | 27/29 | 37/37 | 28/28 | 34/34 | 16/16 | 6/6 | 2/2 | 8/8 | 2/2 | 11/11 | 7/7 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) (N=1) | Part 1: GSK3326595 25mg QD (N=1) | Part 1: GSK3326595 50mg QD (N=1) | Part 1: GSK3326595 100mg QD (N=1) | Part 1: GSK3326595 200mg QD (N=8) | Part 1: GSK3326595 300mg QD (N=3) | Part 1: GSK3326595 400mg QD (N=19) | Part 1: GSK3326595 600mg QD (N=3) | Part 1: GSK3326595 50mg Twice Daily (BID) (N=1) | Part 1: GSK3326595 100mg BID (N=7) | Part 1: GSK3326595 150mg BID (N=6) | Part 1: GSK3326595 200mg BID (N=3) | Part 1: GSK3326595 300mg QD (Food Effect) (N=15) | Part 2: GSK3326595 400mg (TNBC) (N=22) | Part 2: GSK3326595 400mg (mTCC) (N=16) | Part 2: GSK3326595 400mg (GBM) (N=29) | Part 2: GSK3326595 400mg (ER+BC) (N=37) | Part 2: GSK3326595 400mg (HPV+) (N=28) | Part 2: GSK3326595 400mg (ACC) (N=34) | Part 2: GSK3326595 300mg (ACC) (N=16) | Part 2: GSK3326595 400mg (NHL P53 Mutant) (N=6) | Part 2: GSK3326595 300mg (NHL P53 Mutant) (N=2) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) (N=8) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) (N=2) | Part 2: GSK3326595 400mg (NHL P53 Unknown) (N=11) | Part 2: GSK3326595 300mg (NSCLC) (N=7) | Part 3: GSK3326595 100mg + Pembrolizumab 200mg (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (7) | 2 (2) | 2 (2) | 3 (3) | 2 (4) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thalamic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral myocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropsychiatric syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK3326595 12.5 Milligram (mg) Once a Day (QD) (N=1) | Part 1: GSK3326595 25mg QD (N=1) | Part 1: GSK3326595 50mg QD (N=1) | Part 1: GSK3326595 100mg QD (N=1) | Part 1: GSK3326595 200mg QD (N=8) | Part 1: GSK3326595 300mg QD (N=3) | Part 1: GSK3326595 400mg QD (N=19) | Part 1: GSK3326595 600mg QD (N=3) | Part 1: GSK3326595 50mg Twice Daily (BID) (N=1) | Part 1: GSK3326595 100mg BID (N=7) | Part 1: GSK3326595 150mg BID (N=6) | Part 1: GSK3326595 200mg BID (N=3) | Part 1: GSK3326595 300mg QD (Food Effect) (N=15) | Part 2: GSK3326595 400mg (TNBC) (N=22) | Part 2: GSK3326595 400mg (mTCC) (N=16) | Part 2: GSK3326595 400mg (GBM) (N=29) | Part 2: GSK3326595 400mg (ER+BC) (N=37) | Part 2: GSK3326595 400mg (HPV+) (N=28) | Part 2: GSK3326595 400mg (ACC) (N=34) | Part 2: GSK3326595 300mg (ACC) (N=16) | Part 2: GSK3326595 400mg (NHL P53 Mutant) (N=6) | Part 2: GSK3326595 300mg (NHL P53 Mutant) (N=2) | Part 2: GSK3326595 400mg (NHL P53 Wild Type) (N=8) | Part 2: GSK3326595 300mg (NHL P53 Wild Type) (N=2) | Part 2: GSK3326595 400mg (NHL P53 Unknown) (N=11) | Part 2: GSK3326595 300mg (NSCLC) (N=7) | Part 3: GSK3326595 100mg + Pembrolizumab 200mg (N=10)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 10 (13) | 2 (2) | 1 (2) | 2 (2) | 4 (4) | 1 (1) | 12 (15) | 7 (8) | 13 (18) | 11 (19) | 18 (28) | 21 (22) | 22 (27) | 11 (13) | 3 (3) | 0 (0) | 4 (4) | 2 (2) | 4 (4) | 3 (3) | 5 (5)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 5 (8) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 5 (7) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (4) | 2 (3) | 2 (2) | 0 (0) | 5 (5) | 9 (9) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 1 (1) | 9 (9) | 13 (14) | 5 (5) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (4)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 11 (15) | 3 (3) | 0 (0) | 3 (4) | 3 (4) | 1 (2) | 7 (10) | 8 (8) | 9 (12) | 11 (20) | 23 (27) | 16 (19) | 19 (23) | 10 (10) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 4 (4) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (17) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 3 (5) | 1 (1) | 5 (8) | 6 (7) | 14 (18) | 10 (23) | 7 (12) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 4 (5) | 5 (5) | 9 (9) | 5 (6) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (4) | 5 (7) | 3 (3) | 12 (14) | 8 (9) | 7 (9) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 2 (3) | 6 (8) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (5) | 0 (0) | 6 (7) | 4 (4) | 14 (17) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 10 (14) | 0 (0) | 0 (0) | 3 (3) | 3 (5) | 3 (8) | 6 (8) | 11 (14) | 9 (20) | 5 (5) | 13 (15) | 18 (22) | 18 (21) | 9 (17) | 6 (10) | 0 (0) | 1 (1) | 0 (0) | 9 (10) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 5 (5) | 7 (7) | 6 (14) | 7 (7) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 4 (5) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 9 (11) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 5 (5) | 5 (5) | 6 (6) | 4 (5) | 13 (16) | 10 (10) | 18 (24) | 5 (7) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 3 (3) | 5 (6) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 6 (6) | 2 (3) | 13 (15) | 6 (6) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 9 (11) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 1 (2) | 5 (7) | 3 (3) | 5 (6) | 3 (3) | 15 (16) | 8 (9) | 20 (22) | 7 (7) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 5 (5) | 6 (6) | 2 (2) | 12 (12) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (4) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 6 (7) | 1 (1) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 5 (6) | 1 (1) | 5 (5) | 5 (5) | 6 (8) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 3 (5) | 5 (6) | 5 (7) | 2 (2) | 7 (8) | 6 (6) | 13 (14) | 3 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 5 (8) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 3 (4) | 8 (9) | 9 (14) | 0 (0) | 18 (19) | 10 (11) | 12 (16) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 4 (5) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (5) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 9 (9) | 2 (2) | 3 (4) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (16) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (6) | 4 (15) | 7 (9) | 6 (9) | 3 (4) | 2 (2) | 5 (6) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 2 (2) | 1 (1) | 8 (9) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 4 (6) | 4 (8) | 0 (0) | 1 (3) | 4 (7) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 4 (6) | 1 (1) | 2 (7) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (8) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura senile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Data was not available for pharmacokinetic parameters in samples that were out of stability or lost in transit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT02783300/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT02783300/SAP_001.pdf